CLINICAL TRIAL: NCT02561195
Title: A PHASE 2, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLINDED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF TWO 3-DOSE REGIMENS OF A CLOSTRIDIUM DIFFICILE VACCINE IN HEALTHY ADULTS AGED 65 TO 85 YEARS
Brief Title: A Study To Investigate Two 3-dose Schedules Of A Clostridium Difficile Vaccine In Healthy Adults Aged 65 to 85 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B5091009
Record Dates: First submitted 2015-07-09; First posted 2015-09-25 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Clostridium Difficile Associated Disease
Keywords: Clostridium difficile, Vaccine.

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Low-dose C. difficile Vaccine (accelerated schedule) (Experimental)
  Interventions: Biological: Clostridium difficile Vaccine
- High-dose C. difficile Vaccine (accelerated schedule) (Experimental)
  Interventions: Biological: Clostridium difficile Vaccine
- Placebo (accelerated schedule) (Placebo Comparator)
  Interventions: Biological: Placebo
- Low-dose C. difficile Vaccine (non-accelerated schedule) (Experimental)
  Interventions: Biological: Clostridium difficile Vaccine
- High-Dose C. difficile Vaccine (non-accelerated schedule) (Experimental)
  Interventions: Biological: Clostridium difficile Vaccine
- Placebo (non-accelerated schedule) (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Clostridium difficile Vaccine — 0.5 mL intramuscular injection.
  Arms: High-Dose C. difficile Vaccine (non-accelerated schedule); High-dose C. difficile Vaccine (accelerated schedule); Low-dose C. difficile Vaccine (accelerated schedule); Low-dose C. difficile Vaccine (non-accelerated schedule)
Biological: Placebo — 0.5 mL intramuscular injection
  Arms: Placebo (accelerated schedule); Placebo (non-accelerated schedule)

SUMMARY:
This study will investigate a Clostridium difficile vaccine in healthy adults aged 65-85 years. Each subject will initially receive 3 doses of vaccine on 1 of 2 vaccination schedules. The study will assess the safety and tolerability of the vaccine as well as the subjects' immune response to the vaccine. One year after the third dose subjects that did not receive placebo will be randomized to receive a fourth dose. Subjects will be followed for up to 4 years after their third vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* Aged 65 to 85 years

Additional Inclusion Criteria for the extension Stage:

* Receipt of all 3 doses of C difficile vaccine (100 µg or 200 µg antigen dose level) in the original portion of the study.

Exclusion Criteria:

* Proven or suspected prior episode of Clostridium difficile associated diarrhea
* Unstable chronic medical condition
* Disease requiring significant change in therapy or hospitalization for worsening disease within 8 weeks before receipt of study vaccine
* Serious chronic disorders
* Congenital or acquired immunodeficiency disorders
* Rheumatologic disorders or other illnesses requiring chronic treatment with known immunosuppressant medications.
* Active or treated leukemia or lymphoma or bone marrow disorder
* Any contraindication to vaccination or vaccine components including previous anaphylactic reaction to any vaccine or vaccine-related components

Additional Exclusion Criteria for the Extension Stage:

* Subjects originally randomized to placebo during the original portion of the study.
* Subjects who have already completed Visit 9 prior to study unblinding.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Avail Clinical Research, LLC, DeLand, Florida
  - QPS-MRA, LLC (Broward Research Group), Hollywood, Florida
  - QPS-MRA, LLC (Miami Research Associates), South Miami, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Vince & Associates Clinical Research, Inc., Overland Park, Kansas
  - Vince & Associates Clinical Research, Inc, Overland Park, Kansas
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Center of Nevada LLC, Las Vegas, Nevada
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Benchmark Research, Austin, Texas
  - Texas Center For Drug Development, Inc., Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Remich S, Kitchin N, Peterson J, Li P, Pride MW, Brock L, Anderson AS, Gruber WC, Jansen KU, Lockhart SP, Webber C. A Phase 2 Extension Study Evaluating the Immunogenicity, Safety, and Tolerability of 3 or 4 Doses of a Clostridioides difficile Vaccine in Healthy US Adults Aged 65 to 85 Years. J Infect Dis. 2024 Feb 14;229(2):367-375. doi: 10.1093/infdis/jiad307. PMID 37531657
- [Derived] Kitchin N, Remich SA, Peterson J, Peng Y, Gruber WC, Jansen KU, Pride MW, Anderson AS, Knirsch C, Webber C. A Phase 2 Study Evaluating the Safety, Tolerability, and Immunogenicity of Two 3-Dose Regimens of a Clostridium difficile Vaccine in Healthy US Adults Aged 65 to 85 Years. Clin Infect Dis. 2020 Jan 1;70(1):1-10. doi: 10.1093/cid/ciz153. PMID 31125055
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5091009&StudyName=A%20Phase%202%2C%20Placebo-controlled%2C%20Randomized%2C%20Observer-blinded%20Study%20To%20Evaluate%20The%20Safety%2C%20Tolerability%2C%20And%20Immunogenicity%20Of%20Two%203-dose%20Regimens%20Of%20A%20Clostridium%20Difficile%20Vaccine%20In%20Healthy%20Adults%20Aged%2065%20To%2085%20Years

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants initially randomized in the month and day regimens who received the first 3 doses of Clostridium difficile vaccine (100 micro gram (mcg) or 200 mcg) were enrolled into the extension stage.
Groups:
- Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen: Participants received 100 microgram (mcg) of Clostridium difficile vaccine intramuscularly on Day 1, 8 and 30 visits. Participants were followed up to 12 months after the last vaccination.
- Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen: Participants received 200 mcg of Clostridium difficile vaccine intramuscularly on Day 1, 8 and 30 visits. Participants were followed up to 12 months after the last vaccination.
- Placebo: Day 1, 8 and 30 Regimen: Participants received placebo saline intramuscularly on Day 1, 8 and 30 visits. Participants were followed up to 12 months after the last vaccination.
- Clostridium Difficile Vaccine(100 mcg): Month 0, 1 and 6 Regimen: Participants received 100 mcg of Clostridium difficile vaccine intramuscularly at Month 0 (Day 1), 1 and 6 visits. Participants were followed up to 12 months after the third vaccination.
- Clostridium Difficile Vaccine(200 mcg): Month 0, 1 and 6 Regimen: Participants received 200 mcg of Clostridium difficile vaccine intramuscularly at Month 0 (Day 1), 1 and 6 visits. Participants were followed up to 12 months after the last vaccination.
- Placebo: Month 0, 1 and 6 Regimen: Participants received placebo saline intramuscularly at Month 0 (Day 1), 1 and 6 visits. Participants were followed up to 12 months after the last vaccination.
- 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen; 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 100 mcg dose level received placebo intramuscularly as the fourth dose in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
- 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 100 mcg dose level received fourth dose of Clostridium difficile vaccine intramuscularly at the 100 mcg dose level in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
- 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen; 200mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 200 mcg dose level received placebo as the fourth dose in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
- 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen; 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 200 mcg dose level received fourth dose of Clostridium difficile vaccine intramuscularly at the 200 mcg dose level in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
- 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 100 mcg dose level received a fourth dose of Clostridium difficile vaccine intramuscularly at the 100 mcg dose level in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
Period: Vaccination 1 to 3
Arm/Group | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg): Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(200 mcg): Month 0, 1 and 6 Regimen | Placebo: Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Started | 183 | 184 | 61 | 183 | 183 | 61 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 182 | 184 | 61 | 183 | 183 | 61 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 160 | 162 | 55 | 157 | 155 | 51 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 22 | 6 | 26 | 28 | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 5 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 1 | 0 | 4 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No longer willing to participate | 2 | 4 | 0 | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 7 | 3 | 1 | 7 | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 2 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 4 | 2 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension Stage (Vaccination 4)
Arm/Group | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg): Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(200 mcg): Month 0, 1 and 6 Regimen | Placebo: Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Started | 0 | 0 | 0 | 0 | 0 | 0 | 16 (Participants who met predefined eligibility criteria enrolled into extension stage.) | 18 (Participants who met predefined eligibility criteria enrolled into extension stage.) | 24 (Participants who met predefined eligibility criteria enrolled into extension stage.) | 22 (Participants who met predefined eligibility criteria enrolled into extension stage.) | 51 (Participants who met predefined eligibility criteria enrolled into extension stage.) | 52 (Participants who met predefined eligibility criteria enrolled into extension stage.) | 58 (Participants who met predefined eligibility criteria enrolled into extension stage.) | 59 (Participants who met predefined eligibility criteria enrolled into extension stage.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 17 | 21 | 20 | 43 | 45 | 51 | 54
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 8 | 7 | 7 | 5
Not completed — Withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 1
Not completed — No Longer Willing To Participate In Study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of the investigational product and had safety data available.
Groups:
- Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen: Participants received 100 mcg of Clostridium difficile vaccine intramuscularly on Day 1, 8 and 30 visits. Participants were followed up to 12 months after the last vaccination
- Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen: Participants received 100 mcg of Clostridium difficile vaccine intramuscularly at Month 0 (Day 1), 1 and 6 visits. Participants were followed up to 12 months after the third vaccination.
- Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen: Participants received 200 mcg of Clostridium difficile vaccine intramuscularly at Month 0 (Day 1), 1 and 6 visits. Participants were followed up to 12 months after the last vaccination.
- Total: Total of all reporting groups
Arm/Group | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen | Placebo: Month 0, 1 and 6 Regimen | Total
Number analyzed (Participants) | 182 | 184 | 61 | 183 | 183 | 61 | 854
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 182 | 184 | 61 | 183 | 183 | 61 | 854
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 106 | 35 | 93 | 97 | 37 | 461
  Male | 89 | 78 | 26 | 90 | 86 | 24 | 393
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 172 | 168 | 59 | 151 | 157 | 56 | 763
  Race: Black | 6 | 16 | 2 | 16 | 13 | 3 | 56
  Race: Asian | 2 | 0 | 0 | 13 | 10 | 1 | 26
  Race: Other | 2 | 0 | 0 | 3 | 3 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Non-Hispanic | 127 | 143 | 48 | 168 | 172 | 57 | 715
  Ethnicity: Hispanic | 55 | 41 | 13 | 15 | 11 | 4 | 139

OUTCOME MEASURES:

1. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin A at Day 37
Description: Toxin A antibodies (threshold >= 219 neutralization units/mL) were measured using neutralization assay.
Time Frame: Day 37 (7 days after Vaccination 3 of Day 1, 8 and 30 regimen)
Population: Evaluable immunogenicity population: all eligible participants randomized to study, received all 3 study vaccinations to which they were randomized, had at least 1 valid assay result from blood drawn within 7 to 14 days after Vaccination 3 and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 165
percentage of participants | 12.5 [5.2 to 24.1] | 68.4 [60.9 to 75.3] | 85.5 [79.1 to 90.5]

2. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin A at Month 7
Description: Toxin A antibodies (threshold >= 219 neutralization units/mL) were measured using neutralization assay.
Time Frame: Month 7 (1 month after Vaccination 3 of Month 0, 1 and 6 regimen)
Population: Evaluable immunogenicity population: all eligible participants randomized to study, received all 3 study vaccinations to which they were randomized, had at least 1 valid assay result from blood drawn within 20 to 45 days after Vaccination 3 and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants | 1.9 [0.0 to 10.1] | 98.2 [94.7 to 99.6] | 95.6 [91.1 to 98.2]

3. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin B at Day 37
Description: Toxin B antibodies (threshold >= 2586 neutralization units/mL) were measured using neutralization assay.
Time Frame: Day 37 (7 days after Vaccination 3 of Day 1, 8 and 30 regimen)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 165
percentage of participants | 1.8 [0.0 to 9.6] | 29.8 [23.1 to 37.3] | 38.8 [31.3 to 46.7]

4. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin B at Month 7
Description: Toxin B antibodies (threshold >= 2586 neutralization units/mL) were measured using neutralization assay.
Time Frame: Month 7 (1 month after Vaccination 3 of Month 0, 1 and 6 regimen)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants | 7.5 [2.1 to 18.2] | 74.8 [67.5 to 81.3] | 87.3 [81.1 to 92.1]

5. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Both Toxin A and Toxin B at Day 37
Description: Toxin A and B antibodies (threshold >= 219 and 2586 neutralization units/mL) were measured using neutralization assay.
Time Frame: Day 37 (7 days after Vaccination 3 of Day 1, 8 and 30 regimen)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 165
percentage of participants | 0.0 [0.0 to 6.4] | 26.3 [19.9 to 33.6] | 38.8 [31.3 to 46.7]

6. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Both Toxin A and Toxin B at Month 7
Description: Toxin A and B antibodies (threshold >= 219 and 2586 neutralization units/mL) were measured using neutralization assay.
Time Frame: Month 7 (1 month after Vaccination 3 of Month 0, 1 and 6 regimen)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants | 0.0 [0.0 to 6.7] | 74.2 [66.8 to 80.8] | 86.1 [79.7 to 91.1]

7. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants With Local Reactions by Severity Within 7 Days After Vaccination 1
Description: Local reactions included pain at injection site, swelling and redness collected by using an electronic diary (e-diary). Pain was graded as: mild (grade 1) (did not interfere with activity), moderate (grade 2)(interfered with activity), severe (grade 3) (prevented daily activity) and grade 4 (emergency room visit or hospitalization). Redness and swelling were graded as: mild (2.5-5.0 centimeter [cm]), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and grade 4 (necrosis).
Time Frame: within 7 days After Vaccination 1
Population: Safety population: all participants who received at least 1 dose of the investigational product. Here "N (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 61 | 179 | 183
percentage of participants
  Pain: Any | 6.6 [1.8 to 15.9] | 19.0 [13.5 to 25.5] | 15.8 [10.9 to 22.0]
  Pain: Mild | 6.6 [1.8 to 15.9] | 17.9 [12.6 to 24.3] | 14.2 [9.5 to 20.1]
  Pain: Moderate | 0.0 [0.0 to 5.9] | 1.1 [0.1 to 4.0] | 1.6 [0.3 to 4.7]
  Pain: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Pain: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Redness: Any | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 1.1 [0.1 to 3.9]
  Redness: Mild | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 1.1 [0.1 to 3.9]
  Redness: Moderate | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Redness: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Redness: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Swelling: Any | 0.0 [0.0 to 5.9] | 1.1 [0.1 to 4.0] | 1.6 [0.3 to 4.7]
  Swelling: Mild | 0.0 [0.0 to 5.9] | 0.6 [0.0 to 3.1] | 0.5 [0.0 to 3.0]
  Swelling: Moderate | 0.0 [0.0 to 5.9] | 0.6 [0.0 to 3.1] | 1.1 [0.1 to 3.9]
  Swelling: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Swelling: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

8. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants With Local Reactions by Severity Within 14 Days After Vaccination 1
Description: Local reactions included pain at injection site, swelling and redness collected by using an electronic diary (e-diary). Pain was graded as: mild (did not interfere with activity), moderate (interfered with activity), severe (prevented daily activity) and grade 4 (emergency room visit or hospitalization). Redness and swelling were graded as: mild (2.5-5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and grade 4 (necrosis).
Time Frame: within 14 days After Vaccination 1
Population: Safety population: all participants who received at least 1 dose of the investigational product. Here "N" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 61 | 182 | 182
percentage of participants
  Pain: Any | 8.2 [2.7 to 18.1] | 24.2 [18.1 to 31.1] | 19.8 [14.3 to 26.3]
  Pain: Mild | 6.6 [1.8 to 15.9] | 22.0 [16.2 to 28.7] | 19.2 [13.8 to 25.7]
  Pain: Moderate | 1.6 [0.0 to 8.8] | 2.2 [0.6 to 5.5] | 0.0 [0.0 to 2.0]
  Pain: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0]
  Pain: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Redness: Any | 1.6 [0.0 to 8.8] | 1.1 [0.1 to 3.9] | 2.2 [0.6 to 5.5]
  Redness: Mild | 1.6 [0.0 to 8.8] | 0.0 [0.0 to 2.0] | 1.1 [0.1 to 3.9]
  Redness: Moderate | 0.0 [0.0 to 5.9] | 1.1 [0.1 to 3.9] | 0.5 [0.0 to 3.0]
  Redness: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0]
  Redness: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Swelling: Any | 0.0 [0.0 to 5.9] | 1.1 [0.1 to 3.9] | 1.1 [0.1 to 3.9]
  Swelling: Mild | 0.0 [0.0 to 5.9] | 0.5 [0.0 to 3.0] | 0.0 [0.0 to 2.0]
  Swelling: Moderate | 0.0 [0.0 to 5.9] | 0.5 [0.0 to 3.0] | 0.5 [0.0 to 3.0]
  Swelling: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0]
  Swelling: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

9. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants With Local Reactions by Severity Within 14 Days After Vaccination 2
Description: as for outcome 8
Time Frame: within 14 days After Vaccination 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 58 | 180 | 179
percentage of participants
  Pain: Any | 0.0 [0.0 to 6.2] | 31.7 [24.9 to 39.0] | 41.3 [34.0 to 48.9]
  Pain: Mild | 0.0 [0.0 to 6.2] | 25.6 [19.4 to 32.6] | 36.3 [29.3 to 43.8]
  Pain: Moderate | 0.0 [0.0 to 6.2] | 6.1 [3.1 to 10.7] | 4.5 [1.9 to 8.6]
  Pain: Severe | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.6 [0.0 to 3.1]
  Pain: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Redness: Any | 1.7 [0.0 to 9.2] | 4.4 [1.9 to 8.6] | 6.7 [3.5 to 11.4]
  Redness: Mild | 1.7 [0.0 to 9.2] | 1.1 [0.1 to 4.0] | 2.8 [0.9 to 6.4]
  Redness: Moderate | 0.0 [0.0 to 6.2] | 1.7 [0.3 to 4.8] | 1.7 [0.3 to 4.8]
  Redness: Severe | 0.0 [0.0 to 6.2] | 1.7 [0.3 to 4.8] | 2.2 [0.6 to 5.6]
  Redness: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Swelling: Any | 0.0 [0.0 to 6.2] | 3.3 [1.2 to 7.1] | 5.6 [2.7 to 10.0]
  Swelling: Mild | 0.0 [0.0 to 6.2] | 1.1 [0.1 to 4.0] | 3.9 [1.6 to 7.9]
  Swelling: Moderate | 0.0 [0.0 to 6.2] | 0.6 [0.0 to 3.1] | 1.1 [0.1 to 4.0]
  Swelling: Severe | 0.0 [0.0 to 6.2] | 1.7 [0.3 to 4.8] | 0.6 [0.0 to 3.1]
  Swelling: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

10. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants With Local Reactions by Severity Within 14 Days After Vaccination 2
Description: as for outcome 8
Time Frame: within 14 days after Vaccination 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 59 | 176 | 177
percentage of participants
  Pain: Any | 5.1 [1.1 to 14.1] | 27.8 [21.4 to 35.1] | 27.7 [21.2 to 34.9]
  Pain: Mild | 5.1 [1.1 to 14.1] | 23.3 [17.3 to 30.2] | 25.4 [19.2 to 32.5]
  Pain: Moderate | 0.0 [0.0 to 6.1] | 4.5 [2.0 to 8.8] | 1.1 [0.1 to 4.0]
  Pain: Severe | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 1.1 [0.1 to 4.0]
  Pain: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Redness: Any | 0.0 [0.0 to 6.1] | 3.4 [1.3 to 7.3] | 1.1 [0.1 to 4.0]
  Redness: Mild | 0.0 [0.0 to 6.1] | 1.7 [0.4 to 4.9] | 0.6 [0.0 to 3.1]
  Redness: Moderate | 0.0 [0.0 to 6.1] | 1.1 [0.1 to 4.0] | 0.0 [0.0 to 2.1]
  Redness: Severe | 0.0 [0.0 to 6.1] | 0.6 [0.0 to 3.1] | 0.6 [0.0 to 3.1]
  Redness: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Swelling: Any | 0.0 [0.0 to 6.1] | 4.0 [1.6 to 8.0] | 4.0 [1.6 to 8.0]
  Swelling: Mild | 0.0 [0.0 to 6.1] | 2.3 [0.6 to 5.7] | 1.1 [0.1 to 4.0]
  Swelling: Moderate | 0.0 [0.0 to 6.1] | 0.6 [0.0 to 3.1] | 1.7 [0.4 to 4.9]
  Swelling: Severe | 0.0 [0.0 to 6.1] | 1.1 [0.1 to 4.0] | 1.1 [0.1 to 4.0]
  Swelling: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]

11. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants With Local Reactions by Severity Within 14 Days After Vaccination 3
Description: as for outcome 8
Time Frame: within 14 days after Vaccination 3
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 57 | 175 | 171
percentage of participants
  Pain: Any | 3.5 [0.4 to 12.1] | 22.9 [16.9 to 29.8] | 22.2 [16.2 to 29.2]
  Pain: Mild | 3.5 [0.4 to 12.1] | 18.9 [13.4 to 25.5] | 21.1 [15.2 to 27.9]
  Pain: Moderate | 0.0 [0.0 to 6.3] | 4.0 [1.6 to 8.1] | 1.2 [0.1 to 4.2]
  Pain: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Pain: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Redness: Any | 0.0 [0.0 to 6.3] | 2.3 [0.6 to 5.7] | 5.3 [2.4 to 9.8]
  Redness: Mild | 0.0 [0.0 to 6.3] | 1.1 [0.1 to 4.1] | 1.8 [0.4 to 5.0]
  Redness: Moderate | 0.0 [0.0 to 6.3] | 1.1 [0.1 to 4.1] | 3.5 [1.3 to 7.5]
  Redness: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Redness: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Swelling: Any | 0.0 [0.0 to 6.3] | 2.9 [0.9 to 6.5] | 5.3 [2.4 to 9.8]
  Swelling: Mild | 0.0 [0.0 to 6.3] | 2.3 [0.6 to 5.7] | 2.9 [1.0 to 6.7]
  Swelling: Moderate | 0.0 [0.0 to 6.3] | 0.6 [0.0 to 3.1] | 2.3 [0.6 to 5.9]
  Swelling: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Swelling: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]

12. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants With Local Reactions by Severity Within 14 Days After Vaccination 3
Description: as for outcome 8
Time Frame: within 14 days after Vaccination 3
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 54 | 168 | 161
percentage of participants
  Pain: Any | 1.9 [0.0 to 9.9] | 22.0 [16.0 to 29.1] | 26.1 [19.5 to 33.6]
  Pain: Mild | 0.0 [0.0 to 6.6] | 19.6 [13.9 to 26.5] | 21.7 [15.6 to 28.9]
  Pain: Moderate | 1.9 [0.0 to 9.9] | 1.8 [0.4 to 5.1] | 4.3 [1.8 to 8.8]
  Pain: Severe | 0.0 [0.0 to 6.6] | 0.6 [0.0 to 3.3] | 0.0 [0.0 to 2.3]
  Pain: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Redness: Any | 0.0 [0.0 to 6.6] | 4.2 [1.7 to 8.4] | 4.3 [1.8 to 8.8]
  Redness: Mild | 0.0 [0.0 to 6.6] | 3.6 [1.3 to 7.6] | 3.7 [1.4 to 7.9]
  Redness: Moderate | 0.0 [0.0 to 6.6] | 0.6 [0.0 to 3.3] | 0.6 [0.0 to 3.4]
  Redness: Severe | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Redness: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Swelling: Any | 0.0 [0.0 to 6.6] | 2.4 [0.7 to 6.0] | 5.0 [2.2 to 9.6]
  Swelling: Mild | 0.0 [0.0 to 6.6] | 2.4 [0.7 to 6.0] | 4.3 [1.8 to 8.8]
  Swelling: Moderate | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.6 [0.0 to 3.4]
  Swelling: Severe | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Swelling: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]

13. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants With Systemic Events by Severity Within 7 Days After Vaccination 1
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, new or worsening joint pain and were recorded by using an e-diary. Fever was graded as mild (38.0 to 38.4 degree Celsius (C)), moderate (38.5 to 38.9 degree C), severe (39.0 to 40.0 degree C), grade 4 (>40.0 degree C). Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours), severe (required intravenous hydration) and grade 4 (hospitalization for hypotensive shock). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours), severe (>=6 stools in 24 hours) and grade 4 (hospitalization). Headache, fatigue, new or worsening muscle pain and new or worsening joint pain was graded as mild (no interference with activity), moderate (some interference with activity), severe (prevents daily activity) and grade 4 (hospitalization).
Time Frame: within 7 days after Vaccination 1
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 61 | 179 | 183
percentage of participants
  Fever: Any: number analyzed (Participants) | 61 | 178 | 183
  Fever: Any | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.1] | 0.5 [0.0 to 3.0]
  Fever: Mild: number analyzed (Participants) | 61 | 178 | 183
  Fever: Mild | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.1] | 0.5 [0.0 to 3.0]
  Fever: Moderate: number analyzed (Participants) | 61 | 178 | 183
  Fever: Moderate | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.0]
  Fever: Severe: number analyzed (Participants) | 61 | 178 | 183
  Fever: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.0]
  Fever: Grade 4: number analyzed (Participants) | 61 | 178 | 183
  Fever: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.0]
  Vomiting: Any | 0.0 [0.0 to 5.9] | 0.6 [0.0 to 3.1] | 0.5 [0.0 to 3.0]
  Vomiting: Mild | 0.0 [0.0 to 5.9] | 0.6 [0.0 to 3.1] | 0.5 [0.0 to 3.0]
  Vomiting: Moderate | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Vomiting: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Vomiting: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Diarrhea: Any | 13.1 [5.8 to 24.2] | 7.8 [4.3 to 12.8] | 9.3 [5.5 to 14.5]
  Diarrhea: Mild | 11.5 [4.7 to 22.2] | 7.3 [3.9 to 12.1] | 7.7 [4.2 to 12.5]
  Diarrhea: Moderate | 1.6 [0.0 to 8.8] | 0.0 [0.0 to 2.0] | 1.6 [0.3 to 4.7]
  Diarrhea: Severe | 0.0 [0.0 to 5.9] | 0.6 [0.0 to 3.1] | 0.0 [0.0 to 2.0]
  Diarrhea: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Headache: Any | 11.5 [4.7 to 22.2] | 7.3 [3.9 to 12.1] | 11.5 [7.2 to 17.0]
  Headache: Mild | 8.2 [2.7 to 18.1] | 5.6 [2.7 to 10.0] | 7.7 [4.2 to 12.5]
  Headache: Moderate | 3.3 [0.4 to 11.3] | 1.7 [0.3 to 4.8] | 3.8 [1.6 to 7.7]
  Headache: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Headache: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Fatigue: Any | 14.8 [7.0 to 26.2] | 10.6 [6.5 to 16.1] | 18.6 [13.2 to 25.0]
  Fatigue: Mild | 11.5 [4.7 to 22.2] | 7.8 [4.3 to 12.8] | 9.3 [5.5 to 14.5]
  Fatigue: Moderate | 3.3 [0.4 to 11.3] | 2.8 [0.9 to 6.4] | 8.7 [5.1 to 13.8]
  Fatigue: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0]
  Fatigue: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  New or worsening muscle pain: Any | 3.3 [0.4 to 11.3] | 6.7 [3.5 to 11.4] | 8.7 [5.1 to 13.8]
  New or worsening muscle pain: Mild | 1.6 [0.0 to 8.8] | 5.0 [2.3 to 9.3] | 4.4 [1.9 to 8.4]
  New or worsening muscle pain: Moderate | 1.6 [0.0 to 8.8] | 1.7 [0.3 to 4.8] | 4.4 [1.9 to 8.4]
  New or worsening muscle pain: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  New or worsening muscle pain: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  New or worsening joint pain: Any | 1.6 [0.0 to 8.8] | 2.8 [0.9 to 6.4] | 8.7 [5.1 to 13.8]
  New or worsening joint pain: Mild | 1.6 [0.0 to 8.8] | 1.1 [0.1 to 4.0] | 3.8 [1.6 to 7.7]
  New or worsening joint pain: Moderate | 0.0 [0.0 to 5.9] | 1.7 [0.3 to 4.8] | 4.4 [1.9 to 8.4]
  New or worsening joint pain: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0]
  New or worsening joint pain: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

14. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants With Systemic Events by Severity Within 14 Days After Vaccination 1
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, new or worsening joint pain and were recorded by using an e-diary. Fever was graded as mild (38.0 to 38.4 C), moderate (38.5 to 38.9 degree C), severe (39.0 to 40.0 degree C), grade 4 (>40.0 degree C). Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours), severe (required intravenous hydration) and grade 4 (hospitalization for hypotensive shock). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours), severe (>=6 stools in 24 hours) and grade 4 (hospitalization). Headache, fatigue, new or worsening muscle pain and new or worsening joint pain was graded as mild (no interference with activity), moderate (some interference with activity), severe (prevents daily activity) and grade 4 (hospitalization).
Time Frame: within 14 days after Vaccination 1
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 61 | 182 | 182
percentage of participants
  Fever: Any | 0.0 [0.0 to 5.9] | 0.5 [0.0 to 3.0] | 0.0 [0.0 to 2.0]
  Fever: Mild | 0.0 [0.0 to 5.9] | 0.5 [0.0 to 3.0] | 0.0 [0.0 to 2.0]
  Fever: Moderate | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Fever: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Fever: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Vomiting: Any | 1.6 [0.0 to 8.8] | 1.6 [0.3 to 4.7] | 0.5 [0.0 to 3.0]
  Vomiting: Mild | 0.0 [0.0 to 5.9] | 0.5 [0.0 to 3.0] | 0.5 [0.0 to 3.0]
  Vomiting: Moderate | 0.0 [0.0 to 5.9] | 1.1 [0.1 to 3.9] | 0.0 [0.0 to 2.0]
  Vomiting: Severe | 1.6 [0.0 to 8.8] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Vomiting: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Diarrhea: Any | 21.3 [11.9 to 33.7] | 19.8 [14.3 to 26.3] | 19.2 [13.8 to 25.7]
  Diarrhea: Mild | 14.8 [7.0 to 26.2] | 17.0 [11.9 to 23.3] | 13.7 [9.1 to 19.6]
  Diarrhea: Moderate | 4.9 [1.0 to 13.7] | 2.7 [0.9 to 6.3] | 4.4 [1.9 to 8.5]
  Diarrhea: Severe | 1.6 [0.0 to 8.8] | 0.0 [0.0 to 2.0] | 1.1 [0.1 to 3.9]
  Diarrhea: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Headache: Any | 27.9 [17.1 to 40.8] | 15.9 [10.9 to 22.1] | 16.5 [11.4 to 22.7]
  Headache: Mild | 19.7 [10.6 to 31.8] | 10.4 [6.4 to 15.8] | 9.3 [5.5 to 14.5]
  Headache: Moderate | 8.2 [2.7 to 18.1] | 5.5 [2.7 to 9.9] | 6.6 [3.5 to 11.2]
  Headache: Severe | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0]
  Headache: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Fatigue: Any | 31.1 [19.9 to 44.3] | 28.6 [22.1 to 35.7] | 26.9 [20.6 to 34.0]
  Fatigue: Mild | 14.8 [7.0 to 26.2] | 14.8 [10.0 to 20.8] | 12.6 [8.2 to 18.4]
  Fatigue: Moderate | 13.1 [5.8 to 24.2] | 13.2 [8.6 to 19.0] | 13.2 [8.6 to 19.0]
  Fatigue: Severe | 3.3 [0.4 to 11.3] | 0.5 [0.0 to 3.0] | 1.1 [0.1 to 3.9]
  Fatigue: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  New or worsening muscle pain: Any | 9.8 [3.7 to 20.2] | 14.3 [9.5 to 20.2] | 14.8 [10.0 to 20.8]
  New or worsening muscle pain: Mild | 3.3 [0.4 to 11.3] | 8.2 [4.7 to 13.2] | 6.0 [3.1 to 10.6]
  New or worsening muscle pain: Moderate | 6.6 [1.8 to 15.9] | 5.5 [2.7 to 9.9] | 7.7 [4.3 to 12.6]
  New or worsening muscle pain: Severe | 0.0 [0.0 to 5.9] | 0.5 [0.0 to 3.0] | 1.1 [0.1 to 3.9]
  New or worsening muscle pain: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  New or worsening joint pain: Any | 9.8 [3.7 to 20.2] | 9.9 [6.0 to 15.2] | 16.5 [11.4 to 22.7]
  New or worsening joint pain: Mild | 3.3 [0.4 to 11.3] | 5.5 [2.7 to 9.9] | 8.2 [4.7 to 13.2]
  New or worsening joint pain: Moderate | 4.9 [1.0 to 13.7] | 4.4 [1.9 to 8.5] | 7.7 [4.3 to 12.6]
  New or worsening joint pain: Severe | 1.6 [0.0 to 8.8] | 0.0 [0.0 to 2.0] | 0.5 [0.0 to 3.0]
  New or worsening joint pain: Grade 4 | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

15. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants With Systemic Events by Severity Within 14 Days After Vaccination 2
Description: as for outcome 14
Time Frame: within 14 days after Vaccination 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 58 | 180 | 179
percentage of participants
  Fever: Any | 0.0 [0.0 to 6.2] | 0.6 [0.0 to 3.1] | 0.0 [0.0 to 2.0]
  Fever: Mild | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Fever: Moderate | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Fever: Severe | 0.0 [0.0 to 6.2] | 0.6 [0.0 to 3.1] | 0.0 [0.0 to 2.0]
  Fever: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Vomiting: Any | 3.4 [0.4 to 11.9] | 0.0 [0.0 to 2.0] | 1.7 [0.3 to 4.8]
  Vomiting: Mild | 3.4 [0.4 to 11.9] | 0.0 [0.0 to 2.0] | 1.7 [0.3 to 4.8]
  Vomiting: Moderate | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Vomiting: Severe | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Vomiting: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Diarrhea: Any | 10.3 [3.9 to 21.2] | 9.4 [5.6 to 14.7] | 12.3 [7.9 to 18.0]
  Diarrhea: Mild | 6.9 [1.9 to 16.7] | 6.7 [3.5 to 11.4] | 8.9 [5.2 to 14.1]
  Diarrhea: Moderate | 3.4 [0.4 to 11.9] | 2.2 [0.6 to 5.6] | 3.4 [1.2 to 7.2]
  Diarrhea: Severe | 0.0 [0.0 to 6.2] | 0.6 [0.0 to 3.1] | 0.0 [0.0 to 2.0]
  Diarrhea: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Headache: Any | 15.5 [7.3 to 27.4] | 12.2 [7.8 to 17.9] | 13.4 [8.8 to 19.3]
  Headache: Mild | 6.9 [1.9 to 16.7] | 8.3 [4.7 to 13.4] | 7.8 [4.3 to 12.8]
  Headache: Moderate | 8.6 [2.9 to 19.0] | 3.9 [1.6 to 7.8] | 5.6 [2.7 to 10.0]
  Headache: Severe | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Headache: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  Fatigue: Any | 20.7 [11.2 to 33.4] | 17.8 [12.5 to 24.2] | 19.0 [13.5 to 25.5]
  Fatigue: Mild | 6.9 [1.9 to 16.7] | 10.0 [6.0 to 15.3] | 10.6 [6.5 to 16.1]
  Fatigue: Moderate | 10.3 [3.9 to 21.2] | 7.8 [4.3 to 12.7] | 7.8 [4.3 to 12.8]
  Fatigue: Severe | 3.4 [0.4 to 11.9] | 0.0 [0.0 to 2.0] | 0.6 [0.0 to 3.1]
  Fatigue: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  New or worsening muscle pain: Any | 8.6 [2.9 to 19.0] | 10.6 [6.5 to 16.0] | 13.4 [8.8 to 19.3]
  New or worsening muscle pain: Mild | 3.4 [0.4 to 11.9] | 5.0 [2.3 to 9.3] | 8.9 [5.2 to 14.1]
  New or worsening muscle pain: Moderate | 5.2 [1.1 to 14.4] | 5.0 [2.3 to 9.3] | 3.9 [1.6 to 7.9]
  New or worsening muscle pain: Severe | 0.0 [0.0 to 6.2] | 0.6 [0.0 to 3.1] | 0.6 [0.0 to 3.1]
  New or worsening muscle pain: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  New or worsening joint pain: Any | 5.2 [1.1 to 14.4] | 6.1 [3.1 to 10.7] | 7.8 [4.3 to 12.8]
  New or worsening joint pain: Mild | 1.7 [0.0 to 9.2] | 1.7 [0.3 to 4.8] | 6.7 [3.5 to 11.4]
  New or worsening joint pain: Moderate | 3.4 [0.4 to 11.9] | 4.4 [1.9 to 8.6] | 1.1 [0.1 to 4.0]
  New or worsening joint pain: Severe | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]
  New or worsening joint pain: Grade 4 | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 2.0] | 0.0 [0.0 to 2.0]

16. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants With Systemic Events by Severity Within 14 Days After Vaccination 2
Description: as for outcome 14
Time Frame: within 14 days after Vaccination 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 59 | 176 | 177
percentage of participants
  Fever: Any | 0.0 [0.0 to 6.1] | 1.1 [0.1 to 4.0] | 0.6 [0.0 to 3.1]
  Fever: Mild | 0.0 [0.0 to 6.1] | 1.1 [0.1 to 4.0] | 0.6 [0.0 to 3.1]
  Fever: Moderate | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Fever: Severe | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Fever: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Vomiting: Any | 1.7 [0.0 to 9.1] | 1.7 [0.4 to 4.9] | 1.1 [0.1 to 4.0]
  Vomiting: Mild | 1.7 [0.0 to 9.1] | 1.7 [0.4 to 4.9] | 0.6 [0.0 to 3.1]
  Vomiting: Moderate | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.6 [0.0 to 3.1]
  Vomiting: Severe | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Vomiting: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Diarrhea: Any | 18.6 [9.7 to 30.9] | 20.5 [14.8 to 27.2] | 14.1 [9.4 to 20.1]
  Diarrhea: Mild | 10.2 [3.8 to 20.8] | 15.3 [10.4 to 21.5] | 10.2 [6.1 to 15.6]
  Diarrhea: Moderate | 8.5 [2.8 to 18.7] | 4.5 [2.0 to 8.8] | 3.4 [1.3 to 7.2]
  Diarrhea: Severe | 0.0 [0.0 to 6.1] | 0.6 [0.0 to 3.1] | 0.6 [0.0 to 3.1]
  Diarrhea: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Headache: Any | 20.3 [11.0 to 32.8] | 14.8 [9.9 to 20.9] | 15.3 [10.3 to 21.4]
  Headache: Mild | 10.2 [3.8 to 20.8] | 9.1 [5.3 to 14.3] | 9.6 [5.7 to 14.9]
  Headache: Moderate | 10.2 [3.8 to 20.8] | 5.1 [2.4 to 9.5] | 5.6 [2.7 to 10.1]
  Headache: Severe | 0.0 [0.0 to 6.1] | 0.6 [0.0 to 3.1] | 0.0 [0.0 to 2.1]
  Headache: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Fatigue: Any | 18.6 [9.7 to 30.9] | 23.9 [17.8 to 30.9] | 18.1 [12.7 to 24.6]
  Fatigue: Mild | 8.5 [2.8 to 18.7] | 11.9 [7.5 to 17.7] | 6.2 [3.1 to 10.8]
  Fatigue: Moderate | 10.2 [3.8 to 20.8] | 11.4 [7.1 to 17.0] | 11.3 [7.0 to 16.9]
  Fatigue: Severe | 0.0 [0.0 to 6.1] | 0.6 [0.0 to 3.1] | 0.6 [0.0 to 3.1]
  Fatigue: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  New or worsening muscle pain: Any | 8.5 [2.8 to 18.7] | 11.9 [7.5 to 17.7] | 10.2 [6.1 to 15.6]
  New or worsening muscle pain: Mild | 5.5 [1.1 to 14.1] | 6.3 [3.2 to 10.9] | 5.1 [2.4 to 9.4]
  New or worsening muscle pain: Moderate | 3.4 [0.4 to 11.7] | 5.1 [2.4 to 9.5] | 4.5 [2.0 to 8.7]
  New or worsening muscle pain: Severe | 0.0 [0.0 to 6.1] | 0.6 [0.0 to 3.1] | 0.6 [0.0 to 3.1]
  New or worsening muscle pain: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  New or worsening joint pain: Any | 5.1 [1.1 to 14.1] | 8.5 [4.8 to 13.7] | 10.2 [6.1 to 15.6]
  New or worsening joint pain: Mild | 0.0 [0.0 to 6.1] | 6.3 [3.2 to 10.9] | 5.1 [2.4 to 9.4]
  New or worsening joint pain: Moderate | 3.4 [0.4 to 11.7] | 2.3 [0.6 to 5.7] | 5.1 [2.4 to 9.4]
  New or worsening joint pain: Severe | 1.7 [0.0 to 9.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  New or worsening joint pain: Grade 4 | 0.0 [0.0 to 6.1] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]

17. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants With Systemic Events by Severity Within 14 Days After Vaccination 3
Description: as for outcome 14
Time Frame: within 14 days after Vaccination 3
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 57 | 175 | 171
percentage of participants
  Fever: Any | 0.0 [0.0 to 6.3] | 0.6 [0.0 to 3.1] | 1.8 [0.4 to 5.0]
  Fever: Mild | 0.0 [0.0 to 6.3] | 0.6 [0.0 to 3.1] | 1.2 [0.1 to 4.2]
  Fever: Moderate | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.6 [0.0 to 3.2]
  Fever: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Fever: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Vomiting: Any | 1.8 [0.0 to 9.4] | 0.0 [0.0 to 2.1] | 1.2 [0.1 to 4.2]
  Vomiting: Mild | 1.8 [0.0 to 9.4] | 0.0 [0.0 to 2.1] | 1.2 [0.1 to 4.2]
  Vomiting: Moderate | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Vomiting: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Vomiting: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Diarrhea: Any | 14.0 [6.3 to 25.8] | 3.4 [1.3 to 7.3] | 8.2 [4.5 to 13.4]
  Diarrhea: Mild | 8.8 [2.9 to 19.3] | 2.9 [0.9 to 6.5] | 7.0 [3.7 to 11.9]
  Diarrhea: Moderate | 3.5 [0.4 to 12.1] | 0.6 [0.0 to 3.1] | 1.2 [0.1 to 4.2]
  Diarrhea: Severe | 1.8 [0.0 to 9.4] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Diarrhea: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Headache: Any | 10.5 [4.0 to 21.5] | 8.0 [4.4 to 13.1] | 11.7 [7.3 to 17.5]
  Headache: Mild | 8.8 [2.9 to 19.3] | 4.6 [2.0 to 8.8] | 4.1 [1.7 to 8.3]
  Headache: Moderate | 1.8 [0.0 to 9.4] | 3.4 [1.3 to 7.3] | 7.0 [3.7 to 11.9]
  Headache: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.6 [0.0 to 3.2]
  Headache: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  Fatigue: Any | 17.5 [8.7 to 29.9] | 9.7 [5.8 to 15.1] | 12.3 [7.8 to 18.2]
  Fatigue: Mild | 10.5 [4.0 to 21.5] | 4.0 [1.6 to 8.1] | 5.8 [2.8 to 10.5]
  Fatigue: Moderate | 7.0 [1.9 to 17.0] | 5.7 [2.8 to 10.3] | 5.8 [2.8 to 10.5]
  Fatigue: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.6 [0.0 to 3.2]
  Fatigue: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  New or worsening muscle pain: Any | 3.5 [0.4 to 12.1] | 5.1 [2.4 to 9.5] | 8.2 [4.5 to 13.4]
  New or worsening muscle pain: Mild | 3.5 [0.4 to 12.1] | 1.7 [0.4 to 4.9] | 4.7 [2.0 to 9.0]
  New or worsening muscle pain: Moderate | 0.0 [0.0 to 6.3] | 3.4 [1.3 to 7.3] | 3.5 [1.3 to 7.5]
  New or worsening muscle pain: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  New or worsening muscle pain: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  New or worsening joint pain: Any | 5.3 [1.1 to 14.6] | 4.0 [1.6 to 8.1] | 5.8 [2.8 to 10.5]
  New or worsening joint pain: Mild | 1.8 [0.0 to 9.4] | 1.1 [0.1 to 4.1] | 4.7 [2.0 to 9.0]
  New or worsening joint pain: Moderate | 3.5 [0.4 to 12.1] | 2.9 [0.9 to 6.5] | 1.2 [0.1 to 4.2]
  New or worsening joint pain: Severe | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]
  New or worsening joint pain: Grade 4 | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.1]

18. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants With Systemic Events by Severity Within 14 Days After Vaccination 3
Description: as for outcome 14
Time Frame: within 14 days after Vaccination 3
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 54 | 168 | 161
percentage of participants
  Fever: Any | 0.0 [0.0 to 6.6] | 1.2 [0.1 to 4.2] | 0.6 [0.0 to 3.4]
  Fever: Mild | 0.0 [0.0 to 6.6] | 1.2 [0.1 to 4.2] | 0.6 [0.0 to 3.4]
  Fever: Moderate | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Fever: Severe | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Fever: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Vomiting: Any | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 1.2 [0.2 to 4.4]
  Vomiting: Mild | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 1.2 [0.2 to 4.4]
  Vomiting: Moderate | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Vomiting: Severe | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Vomiting: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Diarrhea: Any | 11.1 [4.2 to 22.6] | 16.7 [11.4 to 23.2] | 12.4 [7.8 to 18.5]
  Diarrhea: Mild | 5.6 [1.2 to 15.4] | 11.3 [6.9 to 17.1] | 9.3 [5.3 to 14.9]
  Diarrhea: Moderate | 5.6 [1.2 to 15.4] | 4.8 [2.1 to 9.2] | 3.1 [1.0 to 7.1]
  Diarrhea: Severe | 0.0 [0.0 to 6.6] | 0.6 [0.0 to 3.3] | 0.0 [0.0 to 2.3]
  Diarrhea: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Headache: Any | 18.5 [9.3 to 31.4] | 12.5 [7.9 to 18.5] | 14.3 [9.3 to 20.7]
  Headache: Mild | 13.0 [5.4 to 24.9] | 8.3 [4.6 to 13.6] | 7.5 [3.9 to 12.7]
  Headache: Moderate | 5.6 [1.2 to 15.4] | 3.0 [1.0 to 6.8] | 6.8 [3.5 to 11.9]
  Headache: Severe | 0.0 [0.0 to 6.6] | 1.2 [0.1 to 4.2] | 0.0 [0.0 to 2.3]
  Headache: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Fatigue: Any | 14.8 [6.6 to 27.1] | 20.8 [15.0 to 27.8] | 16.8 [11.4 to 23.5]
  Fatigue: Mild | 1.9 [0.0 to 9.9] | 14.9 [9.9 to 21.2] | 9.3 [5.3 to 14.9]
  Fatigue: Moderate | 11.1 [4.2 to 22.6] | 4.8 [2.1 to 9.2] | 6.8 [3.5 to 11.9]
  Fatigue: Severe | 1.9 [0.0 to 9.9] | 1.2 [0.1 to 4.2] | 0.6 [0.0 to 3.4]
  Fatigue: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  New or worsening muscle pain: Any | 11.1 [4.2 to 22.6] | 8.3 [4.6 to 13.6] | 10.6 [6.3 to 16.4]
  New or worsening muscle pain: Mild | 1.9 [0.0 to 9.9] | 4.2 [1.7 to 8.4] | 5.0 [2.2 to 9.6]
  New or worsening muscle pain: Moderate | 9.3 [3.1 to 20.3] | 4.2 [1.7 to 8.4] | 5.6 [2.6 to 10.3]
  New or worsening muscle pain: Severe | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  New or worsening muscle pain: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  New or worsening joint pain: Any | 11.1 [4.2 to 22.6] | 7.1 [3.7 to 12.1] | 8.1 [4.4 to 13.4]
  New or worsening joint pain: Mild | 5.6 [1.2 to 15.4] | 1.8 [0.4 to 5.1] | 5.0 [2.2 to 9.6]
  New or worsening joint pain: Moderate | 5.6 [1.2 to 15.4] | 4.8 [2.1 to 9.2] | 3.1 [1.0 to 7.1]
  New or worsening joint pain: Severe | 0.0 [0.0 to 6.6] | 0.6 [0.0 to 3.3] | 0.0 [0.0 to 2.3]
  New or worsening joint pain: Grade 4 | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]

19. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose of study drug that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From Vaccination 1 up to 28 days after Vaccination 3 (Day 58)
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 61 | 182 | 184
percentage of participants | 27.9 | 23.6 | 36.4

20. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants With Treatment Emergent Adverse Events (AEs)
Description: as for outcome 19
Time Frame: From Vaccination 1 up to 28 days after Vaccination 3 (Day 208)
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 61 | 183 | 183
percentage of participants | 54.1 | 53.6 | 55.7

21. Primary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants With Treatment Emergent Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; lack of efficacy in an approved indication. Treatment-emergent serious adverse events are events between first dose of study drug and up to 6 months after last dose of study drug that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From Vaccination 1 up to 6 months after Vaccination 3 (Month 7)
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 61 | 182 | 184
percentage of participants | 0.0 | 6.0 | 3.3

22. Primary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants With Treatment Emergent Serious Adverse Events (SAEs)
Description: as for outcome 21
Time Frame: From Vaccination 1 up to 6 months after Vaccination 3 (Month 12)
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 61 | 183 | 183
percentage of participants | 3.3 | 10.4 | 12.0

23. Secondary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin A at Day 1, 8, 15, 30, and Month 2, 4, 7, 13
Description: Toxin A antibodies were measured using neutralization assay.
Time Frame: Day 1, 8, 15, 30 and Month 2, 4, 7, 13
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 165
percentage of participants
  Day 1: number analyzed (Participants) | 56 | 171 | 164
  Day 1 | 0.0 [0.0 to 6.4] | 1.2 [0.1 to 4.2] | 0.6 [0.0 to 3.4]
  Day 8 | 0.0 [0.0 to 6.4] | 4.7 [2.0 to 9.0] | 6.7 [3.4 to 11.6]
  Day 15 | 0.0 [0.0 to 6.4] | 17.0 [11.7 to 23.4] | 25.0 [18.6 to 32.3]
  Day 30 | 0.0 [0.0 to 6.4] | 26.3 [19.9 to 33.6] | 36.6 [29.2 to 44.5]
  Month 2 | 3.6 [0.4 to 12.3] | 61.4 [53.7 to 68.7] | 85.5 [79.1 to 90.5]
  Month 4: number analyzed (Participants) | 55 | 170 | 165
  Month 4 | 1.8 [0.0 to 9.7] | 29.4 [22.7 to 36.9] | 52.4 [44.5 to 60.3]
  Month 7: number analyzed (Participants) | 54 | 166 | 159
  Month 7 | 0.0 [0.0 to 6.6] | 15.1 [10.0 to 21.4] | 31.4 [24.3 to 39.3]
  Month 13: number analyzed (Participants) | 54 | 158 | 155
  Month 13 | 1.9 [0.0 to 9.9] | 10.1 [5.9 to 15.9] | 25.8 [19.1 to 33.4]

24. Secondary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin B at Day 1, 8, 15, 30 and Month 2, 4, 7, 13
Description: Toxin B antibodies were measured using neutralization assay.
Time Frame: Day 1, 8, 15, 30 and Month 2, 4, 7, 13
Population: Evaluable immunogenicity population: All eligible participants randomized to study, received all 3 study vaccinations to which they were randomized, had at least 1 valid assay result from blood drawn within 7 to 14 days after Vaccination 3 and had no major protocol violations. N= number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 164
percentage of participants
  Day 1 | 5.4 [1.1 to 14.9] | 4.7 [2.0 to 9.0] | 3.7 [1.4 to 7.8]
  Day 8 | 3.6 [0.4 to 12.3] | 9.9 [5.9 to 15.4] | 11.5 [7.1 to 17.4]
  Day 15 | 3.6 [0.4 to 12.3] | 30.4 [23.6 to 37.9] | 37.2 [29.8 to 45.1]
  Day 30 | 3.6 [0.4 to 12.3] | 29.8 [23.1 to 37.3] | 37.2 [29.8 to 45.1]
  Month 2 | 1.8 [0.0 to 9.6] | 29.2 [22.5 to 36.7] | 37.0 [29.6 to 44.8]
  Month 4 | 0.0 [0.0 to 6.5] | 26.5 [20.0 to 33.8] | 31.1 [24.1 to 38.8]
  Month 7 | 0.0 [0.0 to 6.6] | 24.1 [17.8 to 31.3] | 26.4 [19.7 to 34.0]
  Month 13 | 1.9 [0.0 to 9.9] | 19.6 [13.7 to 26.7] | 31.0 [23.8 to 38.9]

25. Secondary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Both Toxin A and Toxin B at Day 1, 8, 15, 30 and Month 2, 4, 7, 13
Description: Toxin A and toxin B antibodies were measured using neutralization assay.
Time Frame: Day 1, 8, 15, 30 and Month 2, 4, 7, 13
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 164
percentage of participants
  Day 1 | 0.0 [0.0 to 6.4] | 0.0 [0.0 to 2.1] | 0.0 [0.0 to 2.2]
  Day 8 | 0.0 [0.0 to 6.4] | 3.5 [1.3 to 7.5] | 4.8 [2.1 to 9.3]
  Day 15 | 0.0 [0.0 to 6.4] | 11.7 [7.3 to 17.5] | 18.3 [12.7 to 25.1]
  Day 30 | 0.0 [0.0 to 6.4] | 15.8 [10.7 to 22.1] | 20.7 [14.8 to 27.7]
  Month 2 | 0.0 [0.0 to 6.4] | 24.0 [17.8 to 31.1] | 36.4 [29.0 to 44.2]
  Month 4 | 0.0 [0.0 to 6.5] | 13.5 [8.8 to 19.6] | 24.4 [18.0 to 31.7]
  Month 7 | 0.0 [0.0 to 6.6] | 8.4 [4.7 to 13.7] | 15.7 [10.4 to 22.3]
  Month 13 | 0.0 [0.0 to 6.6] | 6.3 [3.1 to 11.3] | 15.5 [10.2 to 22.2]

26. Secondary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin A at Day 1, 30, 37, 187 and Month 2, 6, 12, 18
Description: Toxin A antibodies were measured using neutralization assay.
Time Frame: Day 1, 30, 37, 187 and Month 2, 6, 12, 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants
  Day 1 | 1.9 [0.0 to 10.1] | 0.6 [0.0 to 3.4] | 1.3 [0.2 to 4.5]
  Day 30: number analyzed (Participants) | 53 | 162 | 157
  Day 30 | 0.0 [0.0 to 6.7] | 17.3 [11.8 to 24.0] | 19.1 [13.3 to 26.1]
  Day 37: number analyzed (Participants) | 53 | 163 | 157
  Day 37 | 1.9 [0.0 to 10.1] | 43.6 [35.8 to 51.5] | 56.7 [48.6 to 64.6]
  Month 2 | 1.9 [0.0 to 10.1] | 41.1 [33.5 to 49.1] | 57.0 [48.9 to 64.6]
  Month 6 | 1.9 [0.0 to 10.1] | 15.3 [10.2 to 21.8] | 20.3 [14.3 to 27.4]
  Day 187: number analyzed (Participants) | 53 | 162 | 158
  Day 187 | 0.0 [0.0 to 6.7] | 80.2 [73.3 to 86.1] | 84.8 [78.2 to 90.0]
  Month 12: number analyzed (Participants) | 51 | 160 | 155
  Month 12 | 2.0 [0.0 to 10.4] | 71.9 [64.2 to 78.7] | 77.4 [70.0 to 83.7]
  Month 18: number analyzed (Participants) | 51 | 154 | 152
  Month 18 | 3.9 [0.5 to 13.5] | 48.7 [40.6 to 56.9] | 53.3 [45.0 to 61.4]

27. Secondary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for for Toxin B at Day 1, 30, 37, 187 and Month 2, 6, 12, 18
Description: Toxin B antibodies were measured using neutralization assay.
Time Frame: Day 1, 30, 37, 187 and Month 2, 6, 12, 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants
  Day 1 | 3.8 [0.5 to 13.0] | 2.5 [0.7 to 6.2] | 4.4 [1.8 to 8.9]
  Day 30: number analyzed (Participants) | 53 | 162 | 157
  Day 30 | 1.9 [0.0 to 10.1] | 25.9 [19.4 to 33.4] | 36.9 [29.4 to 45.0]
  Day 37: number analyzed (Participants) | 53 | 163 | 157
  Day 37 | 3.8 [0.5 to 13.0] | 28.8 [22.0 to 36.4] | 38.2 [30.6 to 46.3]
  Month 2 | 5.7 [1.2 to 15.7] | 28.8 [22.0 to 36.4] | 36.7 [29.2 to 44.7]
  Month 6 | 0.0 [0.0 to 6.7] | 19.6 [13.8 to 26.6] | 27.8 [21.0 to 35.5]
  Day 187: number analyzed (Participants) | 53 | 162 | 158
  Day 187 | 1.9 [0.0 to 10.1] | 58.0 [50.0 to 65.7] | 63.9 [55.9 to 71.4]
  Month 12: number analyzed (Participants) | 51 | 160 | 155
  Month 12 | 5.9 [1.2 to 16.2] | 44.4 [36.5 to 52.4] | 56.8 [48.6 to 64.7]
  Month 18: number analyzed (Participants) | 51 | 154 | 152
  Month 18 | 7.8 [2.2 to 18.9] | 34.4 [27.0 to 42.5] | 47.4 [39.2 to 55.6]

28. Secondary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Both Toxin A and Toxin B at Day 1, 30, 37, 187 and Month 2, 6, 12, 18
Description: Toxin A and toxin B antibodies were measured using neutralization assay.
Time Frame: Day 1, 30, 37, 187 and Month 2, 6, 12, 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants
  Day 1 | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Day 30: number analyzed (Participants) | 53 | 162 | 157
  Day 30 | 0.0 [0.0 to 6.7] | 10.5 [6.2 to 16.3] | 13.4 [8.5 to 19.7]
  Day 37: number analyzed (Participants) | 53 | 163 | 157
  Day 37 | 0.0 [0.0 to 6.7] | 19.6 [13.8 to 26.6] | 27.4 [20.6 to 35.1]
  Month 2 | 1.9 [0.0 to 10.1] | 20.2 [14.4 to 27.2] | 27.8 [21.0 to 35.5]
  Month 6 | 0.0 [0.0 to 6.7] | 10.4 [6.2 to 16.2] | 11.4 [6.9 to 17.4]
  Day 187: number analyzed (Participants) | 53 | 162 | 158
  Day 187 | 0.0 [0.0 to 6.7] | 54.9 [46.9 to 62.8] | 63.3 [55.3 to 70.8]
  Month 12: number analyzed (Participants) | 51 | 160 | 155
  Month 12 | 2.0 [0.0 to 10.4] | 40.6 [32.9 to 48.7] | 50.3 [42.2 to 58.4]
  Month 18: number analyzed (Participants) | 51 | 154 | 152
  Month 18 | 0.0 [0.0 to 7.0] | 26.6 [19.8 to 34.3] | 32.9 [25.5 to 41.0]

29. Secondary Outcome: Day 1, 8 and 30 Regimen: Geometric Mean Concentration of Toxin A Specific Neutralizing Antibody Levels at Day 1, 8, 15, 30, 37 and Month 2, 4, 7, 13
Description: Geometric mean concentration (GMC) of toxin A specific antibody levels was calculated using back transformations of the logarithmically transformed means of assay results. Confidence interval (CI) for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of concentrations.
Time Frame: Day 1, 8, 15, 30, 37 and Month 2, 4, 7, 13
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: neutralization units/mL
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 165
neutralization units/mL
  Day 1: number analyzed (Participants) | 56 | 171 | 164
  Day 1 | 86 [80.4 to 91.3] | 83 [80.4 to 85.2] | 85 [81.8 to 88.5]
  Day 8 | 88 [82.0 to 95.3] | 98 [87.3 to 110.7] | 104 [90.7 to 119.1]
  Day 15: number analyzed (Participants) | 56 | 171 | 164
  Day 15 | 81 [78.1 to 84.5] | 143 [121.3 to 169.1] | 192 [152.9 to 241.5]
  Day 30: number analyzed (Participants) | 56 | 171 | 164
  Day 30 | 89 [82.7 to 96.3] | 168 [141.2 to 200.1] | 230 [186.8 to 282.4]
  Day 37 | 102 [88.4 to 118.7] | 368 [314.6 to 431.4] | 556 [480.0 to 644.2]
  Month 2 | 95 [85.7 to 105.5] | 295 [255.3 to 340.4] | 484 [415.9 to 562.8]
  Month 4: number analyzed (Participants) | 55 | 170 | 164
  Month 4 | 85 [79.0 to 90.6] | 153 [133.8 to 175.7] | 238 [206.5 to 274.1]
  Month 7: number analyzed (Participants) | 54 | 166 | 159
  Month 7 | 81 [78.1 to 84.8] | 118 [105.0 to 133.1] | 166 [143.7 to 191.2]
  Month 13: number analyzed (Participants) | 54 | 158 | 155
  Month 13 | 89 [80.9 to 96.8] | 105 [94.7 to 116.5] | 138 [119.9 to 159.8]

30. Secondary Outcome: Day 1, 8 and 30 Regimen: Geometric Mean Concentration of Toxin B Specific Neutralizing Antibody Levels at Day 1, 8, 15, 30, 37 and Month 2, 4, 7, 13
Description: GMC of toxin B specific antibody levels was calculated using back transformations of the logarithmically transformed means of assay results. CI for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of concentrations.
Time Frame: Day 1, 8, 15, 30, 37 and Month 2, 4, 7, 13
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: neutralization units/mL
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 165
neutralization units/mL
  Day 1: number analyzed (Participants) | 56 | 171 | 164
  Day 1 | 193 [150.5 to 247.2] | 187 [162.8 to 215.4] | 188 [162.5 to 217.8]
  Day 8 | 190 [149.6 to 241.6] | 273 [215.5 to 345.1] | 290 [226.5 to 372.5]
  Day 15: number analyzed (Participants) | 56 | 171 | 164
  Day 15 | 190 [148.7 to 241.7] | 807 [551.7 to 1180.9] | 1091 [720.1 to 1652.9]
  Day 30: number analyzed (Participants) | 56 | 171 | 164
  Day 30 | 211 [152.7 to 292.9] | 705 [498.4 to 997.0] | 1029 [688.4 to 1539.1]
  Day 37 | 180 [142.3 to 227.1] | 728 [520.8 to 1017.4] | 1219 [831.1 to 1787.5]
  Month 2 | 188 [147.0 to 239.3] | 676 [490.0 to 933.6] | 1125 [786.5 to 1608.7]
  Month 4: number analyzed (Participants) | 55 | 170 | 164
  Month 4 | 181 [143.9 to 226.9] | 513 [389.0 to 676.7] | 836 [608.1 to 1150.0]
  Month 7: number analyzed (Participants) | 54 | 166 | 159
  Month 7 | 179 [144.1 to 222.7] | 475 [368.3 to 612.2] | 755 [559.9 to 1018.5]
  Month 13: number analyzed (Participants) | 54 | 158 | 155
  Month 13 | 178 [142.6 to 221.5] | 447 [350.1 to 569.8] | 828 [618.2 to 1110.2]

31. Secondary Outcome: Month 0, 1 and 6 Regimen: Geometric Mean Concentration of Toxin A Specific Neutralizing Antibody Levels at Day 1, 30, 37, 187 and Month 2, 6, 7, 12, 18
Description: GMC of toxin A specific antibody levels was calculated using back transformations of the logarithmically transformed means of assay results. CI for GMC were back transformations of a CI based on the Student t distribution for the mean logarithm of concentrations.
Time Frame: Day 1, 30, 37, 187 and Month 2, 6, 7, 12, 18
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: neutralization units/mL
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
neutralization units/mL
  Day 1 | 83 [78.3 to 88.9] | 85 [82.3 to 88.6] | 87 [83.1 to 91.2]
  Day 30: number analyzed (Participants) | 53 | 162 | 157
  Day 30 | 82 [77.9 to 85.6] | 137 [115.2 to 163.7] | 149 [122.7 to 181.7]
  Day 37: number analyzed (Participants) | 53 | 163 | 157
  Day 37 | 93 [85.1 to 102.6] | 231 [191.6 to 277.3] | 329 [270.6 to 400.2]
  Month 2 | 83 [78.1 to 89.0] | 214 [180.7 to 253.8] | 301 [250.6 to 362.7]
  Month 6 | 84 [79.0 to 89.6] | 115 [101.5 to 129.5] | 136 [116.4 to 158.2]
  Day 187: number analyzed (Participants) | 53 | 162 | 158
  Day 187 | 80 [77.9 to 82.3] | 500 [422.6 to 591.3] | 744 [618.9 to 894.5]
  Month 7 | 90 [81.9 to 99.0] | 1245 [1102.2 to 1405.6] | 1380 [1198.6 to 1589.5]
  Month 12: number analyzed (Participants) | 51 | 160 | 155
  Month 12 | 89 [79.6 to 99.2] | 378 [323.2 to 441.9] | 473 [402.1 to 556.2]
  Month 18: number analyzed (Participants) | 51 | 154 | 152
  Month 18 | 89 [81.5 to 97.8] | 214 [182.1 to 250.7] | 257 [216.0 to 305.2]

32. Secondary Outcome: Month 0, 1 and 6 Regimen: Geometric Mean Concentration of Toxin B Specific Neutralizing Antibody Levels at Day 1, 30, 37, 187 and Month 2, 6, 7, 12, 18
Description: as for outcome 30
Time Frame: Day 1, 30, 37, 187 and Month 2, 6, 7, 12, 18
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: neutralization units/mL
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
neutralization units/mL
  Day 1 | 231 [172.6 to 308.6] | 177 [154.7 to 201.5] | 191 [163.4 to 223.4]
  Day 30: number analyzed (Participants) | 53 | 162 | 157
  Day 30 | 209 [159.1 to 273.9] | 570 [410.2 to 791.1] | 909 [624.3 to 1324.6]
  Day 37: number analyzed (Participants) | 53 | 163 | 157
  Day 37 | 218 [164.7 to 288.6] | 662 [472.4 to 928.0] | 1071 [738.0 to 1553.2]
  Month 2 | 216 [160.7 to 289.4] | 656 [473.1 to 909.0] | 1029 [718.2 to 1473.0]
  Month 6 | 214 [163.4 to 279.8] | 447 [340.7 to 586.7] | 702 [515.4 to 955.2]
  Day 187: number analyzed (Participants) | 53 | 162 | 158
  Day 187 | 199 [155.0 to 255.1] | 2805 [2162.7 to 3636.9] | 4669 [3585.5 to 6079.0]
  Month 7 | 229 [168.0 to 310.9] | 6255 [4971.0 to 7870.5] | 9549 [7691.2 to 11856.0]
  Month 12: number analyzed (Participants) | 51 | 160 | 155
  Month 12 | 247 [174.2 to 349.4] | 1799 [1431.5 to 2260.1] | 2993 [2365.7 to 3786.0]
  Month 18: number analyzed (Participants) | 51 | 154 | 152
  Month 18 | 263 [187.4 to 370.1] | 1248 [970.6 to 1604.0] | 2178 [1661.6 to 2856.1]

33. Secondary Outcome: Day 1, 8 and 30 Regimen: Geometric Mean Fold Rise in Toxin A Specific Neutralizing Antibody Levels From Baseline at Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Description: Geometric mean fold rise (GMFR) in toxin A specific antibody levels was calculated using back transformations of the logarithmically transformed means of fold rise from baseline with assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise.
Time Frame: Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 165
fold rise
  Day 8: number analyzed (Participants) | 56 | 171 | 164
  Day 8 | 1.03 [0.95 to 1.13] | 1.19 [1.06 to 1.33] | 1.22 [1.07 to 1.40]
  Day 15: number analyzed (Participants) | 56 | 171 | 163
  Day 15 | 0.95 [0.89 to 1.01] | 1.73 [1.47 to 2.04] | 2.27 [1.80 to 2.86]
  Day 30: number analyzed (Participants) | 56 | 171 | 163
  Day 30 | 1.04 [0.95 to 1.14] | 2.03 [1.71 to 2.41] | 2.72 [2.20 to 3.35]
  Day 37: number analyzed (Participants) | 56 | 171 | 164
  Day 37 | 1.20 [1.03 to 1.39] | 4.45 [3.81 to 5.20] | 6.56 [5.65 to 7.62]
  Month 2: number analyzed (Participants) | 56 | 171 | 164
  Month 2 | 1.11 [0.99 to 1.25] | 3.56 [3.09 to 4.10] | 5.71 [4.89 to 6.67]
  Month 4: number analyzed (Participants) | 55 | 170 | 163
  Month 4 | 0.99 [0.91 to 1.06] | 1.85 [1.62 to 2.12] | 2.81 [2.44 to 3.25]
  Month 7: number analyzed (Participants) | 54 | 166 | 158
  Month 7 | 0.95 [0.89 to 1.01] | 1.43 [1.27 to 1.60] | 1.95 [1.68 to 2.26]
  Month 13: number analyzed (Participants) | 54 | 158 | 154
  Month 13 | 1.03 [0.92 to 1.15] | 1.26 [1.14 to 1.40] | 1.64 [1.42 to 1.90]

34. Secondary Outcome: Day 1, 8 and 30 Regimen: Geometric Mean Fold Rise in Toxin B Specific Neutralizing Antibody Levels From Baseline at Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Description: GMFR in toxin B specific antibody levels was calculated using back transformations of the logarithmically transformed means of fold rise from baseline with assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise.
Time Frame: Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Population: Evaluable immunogenicity population: all eligible participants randomized to study, received all 3 study vaccinations to which they were randomized, had at least 1 valid assay result from blood drawn within 7 to 14 days after Vaccination 3 and had no major protocol violations. Here, N= number of participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 164
fold rise
  Day 8 | 0.99 [0.94 to 1.04] | 1.46 [1.24 to 1.72] | 1.55 [1.31 to 1.84]
  Day 15: number analyzed (Participants) | 56 | 171 | 163
  Day 15 | 0.98 [0.94 to 1.03] | 4.31 [3.17 to 5.87] | 5.86 [4.07 to 8.43]
  Day 30: number analyzed (Participants) | 56 | 171 | 163
  Day 30 | 1.10 [0.86 to 1.39] | 3.76 [2.87 to 4.94] | 5.53 [3.89 to 7.85]
  Day 37 | 0.93 [0.84 to 1.04] | 3.89 [2.99 to 5.05] | 6.57 [4.74 to 9.10]
  Month 2 | 0.97 [0.90 to 1.05] | 3.61 [2.82 to 4.63] | 6.06 [4.50 to 8.15]
  Month 4: number analyzed (Participants) | 55 | 170 | 163
  Month 4 | 0.93 [0.84 to 1.02] | 2.73 [2.23 to 3.35] | 4.55 [3.53 to 5.86]
  Month 7: number analyzed (Participants) | 54 | 166 | 158
  Month 7 | 0.96 [0.88 to 1.04] | 2.52 [2.09 to 3.03] | 4.05 [3.20 to 5.12]
  Month 13: number analyzed (Participants) | 54 | 158 | 154
  Month 13 | 0.95 [0.87 to 1.04] | 2.40 [2.00 to 2.89] | 4.44 [3.46 to 5.69]

35. Secondary Outcome: Month 0, 1 and 6 Regimen: Geometric Mean Fold Rise in Toxin A Specific Neutralizing Antibody Levels From Baseline at Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Description: GMFR in toxin A specific antibody levels was calculated using back transformations of the logarithmically transformed means of fold rise from baseline with assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise.
Time Frame: Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
fold rise
  Day 30: number analyzed (Participants) | 53 | 162 | 157
  Day 30 | 0.98 [0.90 to 1.06] | 1.61 [1.35 to 1.91] | 1.71 [1.41 to 2.09]
  Day 37: number analyzed (Participants) | 53 | 163 | 157
  Day 37 | 1.12 [0.99 to 1.26] | 2.70 [2.25 to 3.24] | 3.78 [3.10 to 4.59]
  Month 2 | 1.00 [0.91 to 1.10] | 2.51 [2.12 to 2.97] | 3.46 [2.88 to 4.16]
  Month 6 | 1.01 [0.92 to 1.11] | 1.34 [1.19 to 1.52] | 1.56 [1.34 to 1.81]
  Day 187: number analyzed (Participants) | 53 | 162 | 158
  Day 187 | 0.96 [0.89 to 1.03] | 5.85 [4.92 to 6.95] | 8.54 [7.08 to 10.30]
  Month 7 | 1.08 [0.96 to 1.22] | 14.58 [12.82 to 16.58] | 15.85 [13.70 to 18.34]
  Month 12: number analyzed (Participants) | 51 | 160 | 155
  Month 12 | 1.06 [0.93 to 1.21] | 4.42 [3.77 to 5.19] | 5.45 [4.62 to 6.42]
  Month 18: number analyzed (Participants) | 51 | 154 | 152
  Month 18 | 1.07 [0.95 to 1.20] | 2.51 [2.14 to 2.95] | 2.95 [2.49 to 3.50]

36. Secondary Outcome: Month 0, 1 and 6 Regimen: Geometric Mean Fold Rise in Toxin B Specific Neutralizing Antibody Levels From Baseline at Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Description: GMFR for toxin B specific antibody levels was calculated using back transformations of the logarithmically transformed means of fold rise from baseline with assay results. CI for GMFR were back transformations of a CI based on the Student t distribution for the mean logarithm of the mean fold rise.
Time Frame: Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
fold rise
  Day 30: number analyzed (Participants) | 53 | 162 | 157
  Day 30 | 0.90 [0.74 to 1.10] | 3.28 [2.48 to 4.35] | 4.75 [3.47 to 6.50]
  Day 37: number analyzed (Participants) | 53 | 163 | 157
  Day 37 | 0.94 [0.79 to 1.13] | 3.75 [2.85 to 4.94] | 5.59 [4.16 to 7.51]
  Month 2 | 0.93 [0.74 to 1.18] | 3.71 [2.83 to 4.87] | 5.38 [4.05 to 7.15]
  Month 6 | 0.93 [0.76 to 1.13] | 2.53 [2.06 to 3.12] | 3.67 [2.90 to 4.65]
  Day 187: number analyzed (Participants) | 53 | 162 | 158
  Day 187 | 0.86 [0.72 to 1.03] | 15.85 [12.54 to 20.05] | 24.44 [19.14 to 31.20]
  Month 7 | 0.99 [0.81 to 1.21] | 35.43 [28.35 to 44.27] | 49.98 [40.24 to 62.07]
  Month 12: number analyzed (Participants) | 51 | 160 | 155
  Month 12 | 1.04 [0.84 to 1.30] | 10.19 [8.32 to 12.49] | 15.54 [12.61 to 19.13]
  Month 18: number analyzed (Participants) | 51 | 154 | 152
  Month 18 | 1.11 [0.90 to 1.39] | 7.07 [5.69 to 8.77] | 11.21 [8.85 to 14.21]

37. Secondary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Toxin A Specific Antibody Levels at Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Description: Toxin A antibodies were measured using neutralization assay.
Time Frame: Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 164
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 6.4] | 3.5 [1.3 to 7.5] | 4.9 [2.1 to 9.4]
  Day 8: >=8 fold rise | 0.0 [0.0 to 6.4] | 2.9 [1.0 to 6.7] | 4.3 [1.7 to 8.6]
  Day 8: >=16 fold rise | 0.0 [0.0 to 6.4] | 2.3 [0.6 to 5.9] | 3.0 [1.0 to 7.0]
  Day 8: >=32 fold rise | 0.0 [0.0 to 6.4] | 2.3 [0.6 to 5.9] | 2.4 [0.7 to 6.1]
  Day 15: >=4 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=4 fold rise | 0.0 [0.0 to 6.4] | 14.6 [9.7 to 20.8] | 19.6 [13.8 to 26.6]
  Day 15: >=8 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=8 fold rise | 0.0 [0.0 to 6.4] | 9.9 [5.9 to 15.4] | 17.8 [12.3 to 24.5]
  Day 15: >=16 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=16 fold rise | 0.0 [0.0 to 6.4] | 5.8 [2.8 to 10.5] | 14.1 [9.2 to 20.4]
  Day 15: >=32 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=32 fold rise | 0.0 [0.0 to 6.4] | 4.7 [2.0 to 9.0] | 9.2 [5.2 to 14.7]
  Day 30: >=4 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=4 fold rise | 0.0 [0.0 to 6.4] | 17.5 [12.2 to 24.1] | 25.8 [19.2 to 33.2]
  Day 30: >=8 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=8 fold rise | 0.0 [0.0 to 6.4] | 8.2 [4.5 to 13.4] | 17.2 [11.7 to 23.9]
  Day 30: >=16 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=16 fold rise | 0.0 [0.0 to 6.4] | 5.8 [2.8 to 10.5] | 13.5 [8.7 to 19.7]
  Day 30: >=32 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=32 fold rise | 0.0 [0.0 to 6.4] | 5.3 [2.4 to 9.8] | 8.6 [4.8 to 14.0]
  Day 37: >=4 fold rise | 5.4 [1.1 to 14.9] | 46.8 [39.1 to 54.6] | 65.2 [57.4 to 72.5]
  Day 37: >=8 fold rise | 0.0 [0.0 to 6.4] | 25.1 [18.8 to 32.3] | 40.9 [33.3 to 48.8]
  Day 37: >=16 fold rise | 0.0 [0.0 to 6.4] | 8.8 [5.0 to 14.1] | 14.0 [9.1 to 20.3]
  Day 37: >=32 fold rise | 0.0 [0.0 to 6.4] | 3.5 [1.3 to 7.5] | 8.5 [4.7 to 13.9]
  Month 2: >=4 fold rise | 1.8 [0.0 to 9.6] | 32.7 [25.8 to 40.3] | 59.1 [51.2 to 66.7]
  Month 2: >=8 fold rise | 0.0 [0.0 to 6.4] | 18.1 [12.7 to 24.7] | 31.1 [24.1 to 38.8]
  Month 2: >=16 fold rise | 0.0 [0.0 to 6.4] | 5.8 [2.8 to 10.5] | 12.8 [8.1 to 18.9]
  Month 2: >=32 fold rise | 0.0 [0.0 to 6.4] | 3.5 [1.3 to 7.5] | 6.7 [3.4 to 11.7]
  Month 4: >=4 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=4 fold rise | 0.0 [0.0 to 6.5] | 13.5 [8.8 to 19.6] | 24.5 [18.1 to 31.9]
  Month 4: >=8 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=8 fold rise | 0.0 [0.0 to 6.5] | 7.1 [3.7 to 12.0] | 12.9 [8.2 to 19.0]
  Month 4: >=16 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=16 fold rise | 0.0 [0.0 to 6.5] | 4.1 [1.7 to 8.3] | 5.5 [2.6 to 10.2]
  Month 4: >=32 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=32 fold rise | 0.0 [0.0 to 6.5] | 1.2 [0.1 to 4.2] | 2.5 [0.7 to 6.2]
  Month 7: >=4 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=4 fold rise | 0.0 [0.0 to 6.6] | 9.0 [5.1 to 14.5] | 16.5 [11.0 to 23.2]
  Month 7: >=8 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=8 fold rise | 0.0 [0.0 to 6.6] | 5.4 [2.5 to 10.0] | 10.1 [5.9 to 15.9]
  Month 7: >=16 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=16 fold rise | 0.0 [0.0 to 6.6] | 1.8 [0.4 to 5.2] | 5.7 [2.6 to 10.5]
  Month 7: >=32 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=32 fold rise | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.2] | 1.3 [0.2 to 4.5]
  Month 13: >=4 fold rise: number analyzed (Participants) | 56 | 158 | 154
  Month 13: >=4 fold rise | 1.9 [0.0 to 9.9] | 6.3 [3.1 to 11.3] | 16.2 [10.8 to 23.0]
  Month 13: >=8 fold rise: number analyzed (Participants) | 56 | 158 | 154
  Month 13: >=8 fold rise | 0.0 [0.0 to 6.6] | 3.8 [1.4 to 8.1] | 9.7 [5.6 to 15.6]
  Month 13: >=16 fold rise: number analyzed (Participants) | 56 | 158 | 154
  Month 13: >=16 fold rise | 0.0 [0.0 to 6.6] | 0.6 [0.0 to 3.5] | 3.2 [1.1 to 7.4]
  Month 13: >=32 fold rise: number analyzed (Participants) | 56 | 158 | 154
  Month 13: >=32 fold rise | 0.0 [0.0 to 6.6] | 0.6 [0.0 to 3.5] | 0.6 [0.0 to 3.6]

38. Secondary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Toxin B Specific Antibody Levels at Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Description: Toxin B antibodies were measured using neutralization assay.
Time Frame: Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 164
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 6.4] | 11.7 [7.3 to 17.5] | 14.6 [9.6 to 21.0]
  Day 8: >=8 fold rise | 0.0 [0.0 to 6.4] | 8.2 [4.5 to 13.4] | 8.5 [4.7 to 13.9]
  Day 8: >=16 fold rise | 0.0 [0.0 to 6.4] | 4.7 [2.0 to 9.0] | 4.9 [2.1 to 9.4]
  Day 8: >=32 fold rise | 0.0 [0.0 to 6.4] | 3.5 [1.3 to 7.5] | 3.0 [1.0 to 7.0]
  Day 15: >=4 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=4 fold rise | 0.0 [0.0 to 6.4] | 36.8 [29.6 to 44.5] | 41.1 [33.5 to 49.1]
  Day 15: >=8 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=8 fold rise | 0.0 [0.0 to 6.4] | 33.3 [26.3 to 40.9] | 38.7 [31.1 to 46.6]
  Day 15: >=16 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=16 fold rise | 0.0 [0.0 to 6.4] | 26.3 [19.9 to 33.6] | 35.0 [27.7 to 42.8]
  Day 15: >=32 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=32 fold rise | 0.0 [0.0 to 6.4] | 20.5 [14.7 to 27.3] | 29.4 [22.6 to 37.1]
  Day 30: >=4 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=4 fold rise | 1.8 [0.0 to 9.6] | 39.2 [31.8 to 46.9] | 42.3 [34.6 to 50.3]
  Day 30: >=8 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=8 fold rise | 1.8 [0.0 to 9.6] | 33.3 [26.3 to 40.9] | 39.9 [32.3 to 47.8]
  Day 30: >=16 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=16 fold rise | 1.8 [0.0 to 9.6] | 22.8 [16.7 to 29.8] | 37.4 [30.0 to 45.3]
  Day 30: >=32 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=32 fold rise | 1.8 [0.0 to 9.6] | 17.0 [11.7 to 23.4] | 27.6 [20.9 to 35.1]
  Day 37: >=4 fold rise | 0.0 [0.0 to 6.4] | 41.5 [34.0 to 49.3] | 46.3 [38.5 to 54.3]
  Day 37: >=8 fold rise | 0.0 [0.0 to 6.4] | 33.9 [26.9 to 41.5] | 40.2 [32.7 to 48.2]
  Day 37: >=16 fold rise | 0.0 [0.0 to 6.4] | 24.0 [17.8 to 31.1] | 37.2 [29.8 to 45.1]
  Day 37: >=32 fold rise | 0.0 [0.0 to 6.4] | 16.4 [11.2 to 22.8] | 27.4 [20.8 to 34.9]
  Month 2: >=4 fold rise | 0.0 [0.0 to 6.4] | 39.2 [31.8 to 46.9] | 46.3 [38.5 to 54.3]
  Month 2: >=8 fold rise | 0.0 [0.0 to 6.4] | 32.2 [25.2 to 39.7] | 38.4 [30.9 to 46.3]
  Month 2: >=16 fold rise | 0.0 [0.0 to 6.4] | 22.8 [16.7 to 29.8] | 34.1 [26.9 to 41.9]
  Month 2: >=32 fold rise | 0.0 [0.0 to 6.4] | 14.6 [9.7 to 20.8] | 24.4 [18.0 to 31.7]
  Month 4: >=4 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=4 fold rise | 0.0 [0.0 to 6.5] | 35.9 [28.7 to 43.6] | 42.3 [34.6 to 50.3]
  Month 4: >=8 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=8 fold rise | 0.0 [0.0 to 6.5] | 23.5 [17.4 to 30.6] | 34.4 [27.1 to 42.2]
  Month 4: >=16 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=16 fold rise | 0.0 [0.0 to 6.5] | 14.7 [9.7 to 20.9] | 25.8 [19.2 to 33.2]
  Month 4: >=32 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=32 fold rise | 0.0 [0.0 to 6.5] | 5.9 [2.9 to 10.6] | 16.6 [11.2 to 23.2]
  Month 7: >=4 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=4 fold rise | 0.0 [0.0 to 6.6] | 34.9 [27.7 to 42.7] | 45.6 [37.6 to 53.7]
  Month 7: >=8 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=8 fold rise | 0.0 [0.0 to 6.6] | 19.9 [14.1 to 26.8] | 30.4 [23.3 to 38.2]
  Month 7: >=16 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=16 fold rise | 0.0 [0.0 to 6.6] | 8.4 [4.7 to 13.7] | 20.3 [14.3 to 27.4]
  Month 7: >=32 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=32 fold rise | 0.0 [0.0 to 6.6] | 1.8 [0.4 to 5.2] | 13.3 [8.4 to 19.6]
  Month 13: >=4 fold rise: number analyzed (Participants) | 54 | 158 | 154
  Month 13: >=4 fold rise | 0.0 [0.0 to 6.6] | 35.4 [28.0 to 43.4] | 46.8 [38.7 to 55.0]
  Month 13: >=8 fold rise: number analyzed (Participants) | 54 | 158 | 154
  Month 13: >=8 fold rise | 0.0 [0.0 to 6.6] | 17.7 [12.1 to 24.6] | 30.5 [23.4 to 38.4]
  Month 13: >=16 fold rise: number analyzed (Participants) | 54 | 158 | 154
  Month 13: >=16 fold rise | 0.0 [0.0 to 6.6] | 10.8 [6.4 to 16.7] | 20.8 [14.7 to 28.0]
  Month 13: >=32 fold rise: number analyzed (Participants) | 54 | 158 | 154
  Month 13: >=32 fold rise | 0.0 [0.0 to 6.6] | 1.3 [0.2 to 4.5] | 14.9 [9.7 to 21.6]

39. Secondary Outcome: Day 1, 8 and 30 Regimen: Percentage of Participants Achieving>=4,>=8,>=16,>=32 Fold Rise From Baseline in Both Toxin A and Toxin B Specific Antibody Levels at Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Description: Toxin A and toxin B antibodies were measured using neutralization assay.
Time Frame: Day 8, 15, 30, 37 and Month 2, 4, 7, 13
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 56 | 171 | 164
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 6.4] | 3.5 [1.3 to 7.5] | 3.0 [1.0 to 7.0]
  Day 8: >=8 fold rise | 0.0 [0.0 to 6.4] | 2.9 [1.0 to 6.7] | 1.8 [0.4 to 5.3]
  Day 8: >=16 fold rise | 0.0 [0.0 to 6.4] | 2.3 [0.6 to 5.9] | 1.2 [0.1 to 4.3]
  Day 8: >=32 fold rise | 0.0 [0.0 to 6.4] | 1.8 [0.4 to 5.0] | 0.6 [0.0 to 3.4]
  Day 15: >=4 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=4 fold rise | 0.0 [0.0 to 6.4] | 12.3 [7.8 to 18.2] | 17.2 [11.7 to 23.9]
  Day 15: >=8 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=8 fold rise | 0.0 [0.0 to 6.4] | 7.6 [4.1 to 12.6] | 14.7 [9.7 to 21.1]
  Day 15: >=16 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=16 fold rise | 0.0 [0.0 to 6.4] | 4.7 [2.0 to 9.0] | 9.8 [5.7 to 15.5]
  Day 15: >=32 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 15: >=32 fold rise | 0.0 [0.0 to 6.4] | 3.5 [1.3 to 7.5] | 4.9 [2.1 to 9.4]
  Day 30: >=4 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=4 fold rise | 0.0 [0.0 to 6.4] | 13.5 [8.7 to 19.5] | 20.2 [14.4 to 27.2]
  Day 30: >=8 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=8 fold rise | 0.0 [0.0 to 6.4] | 7.0 [3.7 to 11.9] | 14.1 [9.2 to 20.4]
  Day 30: >=16 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=16 fold rise | 0.0 [0.0 to 6.4] | 4.1 [1.7 to 8.3] | 11.0 [6.7 to 16.9]
  Day 30: >=32 fold rise: number analyzed (Participants) | 56 | 171 | 163
  Day 30: >=32 fold rise | 0.0 [0.0 to 6.4] | 3.5 [1.3 to 7.5] | 5.5 [2.6 to 10.2]
  Day 37: >=4 fold rise | 0.0 [0.0 to 6.4] | 25.1 [18.8 to 32.3] | 36.0 [28.6 to 43.8]
  Day 37: >=8 fold rise | 0.0 [0.0 to 6.4] | 14.6 [9.7 to 20.8] | 25.6 [19.1 to 33.0]
  Day 37: >=16 fold rise | 0.0 [0.0 to 6.4] | 6.4 [3.3 to 11.2] | 11.6 [7.1 to 17.5]
  Day 37: >=32 fold rise | 0.0 [0.0 to 6.4] | 2.3 [0.6 to 5.9] | 6.7 [3.4 to 11.7]
  Month 2: >=4 fold rise | 0.0 [0.0 to 6.4] | 21.6 [15.7 to 28.6] | 34.8 [27.5 to 42.6]
  Month 2: >=8 fold rise | 0.0 [0.0 to 6.4] | 11.7 [7.3 to 17.5] | 21.3 [15.3 to 28.4]
  Month 2: >=16 fold rise | 0.0 [0.0 to 6.4] | 2.9 [1.0 to 6.7] | 10.4 [6.2 to 16.1]
  Month 2: >=32 fold rise | 0.0 [0.0 to 6.4] | 2.3 [0.6 to 5.9] | 5.5 [2.5 to 10.2]
  Month 4: >=4 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=4 fold rise | 0.0 [0.0 to 6.5] | 8.8 [5.0 to 14.1] | 19.0 [13.3 to 25.9]
  Month 4: >=8 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=8 fold rise | 0.0 [0.0 to 6.5] | 4.1 [1.7 to 8.3] | 9.2 [5.2 to 14.7]
  Month 4: >=16 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=16 fold rise | 0.0 [0.0 to 6.5] | 2.4 [0.6 to 5.9] | 3.1 [1.0 to 7.0]
  Month 4: >=32 fold rise: number analyzed (Participants) | 55 | 170 | 163
  Month 4: >=32 fold rise | 0.0 [0.0 to 6.5] | 0.6 [0.0 to 3.2] | 1.2 [0.1 to 4.4]
  Month 7: >=4 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=4 fold rise | 0.0 [0.0 to 6.6] | 7.2 [3.8 to 12.3] | 13.9 [8.9 to 20.3]
  Month 7: >=8 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=8 fold rise | 0.0 [0.0 to 6.6] | 3.6 [1.3 to 7.7] | 7.0 [3.5 to 12.1]
  Month 7: >=16 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=16 fold rise | 0.0 [0.0 to 6.6] | 0.6 [0.0 to 3.3] | 3.2 [1.0 to 7.2]
  Month 7: >=32 fold rise: number analyzed (Participants) | 54 | 166 | 158
  Month 7: >=32 fold rise | 0.0 [0.0 to 0.6] | 0.0 [0.0 to 2.2] | 0.0 [0.0 to 2.3]
  Month 13: >=4 fold rise: number analyzed (Participants) | 54 | 158 | 154
  Month 13: >=4 fold rise | 0.0 [0.0 to 6.6] | 5.1 [2.2 to 9.7] | 14.3 [9.2 to 20.8]
  Month 13: >=8 fold rise: number analyzed (Participants) | 54 | 158 | 154
  Month 13: >=8 fold rise | 0.0 [0.0 to 6.6] | 2.5 [0.7 to 6.4] | 6.5 [3.2 to 11.6]
  Month 13: >=16 fold rise: number analyzed (Participants) | 54 | 158 | 154
  Month 13: >=16 fold rise | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.3] | 1.3 [0.2 to 4.6]
  Month 13: >=32 fold rise: number analyzed (Participants) | 54 | 158 | 154
  Month 13: >=32 fold rise | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 2.3] | 0.0 [0.0 to 2.4]

40. Secondary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Toxin A Specific Antibody Levels at Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Description: Toxin A antibodies were measured using neutralization assay.
Time Frame: Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants
  Day 30: >=4 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=4 fold rise | 0.0 [0.0 to 6.7] | 14.2 [9.2 to 20.5] | 14.0 [9.0 to 20.4]
  Day 30: >=8 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=8 fold rise | 0.0 [0.0 to 6.7] | 12.3 [7.7 to 18.4] | 11.5 [6.9 to 17.5]
  Day 30: >=16 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=16 fold rise | 0.0 [0.0 to 6.7] | 6.8 [3.4 to 11.8] | 10.2 [5.9 to 16.0]
  Day 30: >=32 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=32 fold rise | 0.0 [0.0 to 6.7] | 2.5 [0.7 to 6.2] | 6.4 [3.1 to 11.4]
  Day 37: >=4 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=4 fold rise | 0.0 [0.0 to 6.7] | 28.2 [21.5 to 35.8] | 40.1 [32.4 to 48.2]
  Day 37: >=8 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=8 fold rise | 0.0 [0.0 to 6.7] | 16.0 [10.7 to 22.5] | 26.8 [20.0 to 34.4]
  Day 37: >=16 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=16 fold rise | 0.0 [0.0 to 6.7] | 6.1 [3.0 to 11.0] | 12.7 [8.0 to 19.0]
  Day 37: >=32 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=32 fold rise | 0.0 [0.0 to 6.7] | 3.1 [1.0 to 7.0] | 7.0 [3.5 to 12.2]
  Month 2: >=4 fold rise | 1.9 [0.0 to 10.1] | 28.2 [21.5 to 35.8] | 36.1 [28.6 to 44.1]
  Month 2: >=8 fold rise | 0.0 [0.0 to 6.7] | 14.7 [9.7 to 21.1] | 21.5 [15.4 to 28.8]
  Month 2: >=16 fold rise | 0.0 [0.0 to 6.7] | 6.7 [3.4 to 11.8] | 12.0 [7.4 to 18.1]
  Month 2: >=32 fold rise | 0.0 [0.0 to 6.7] | 2.5 [0.7 to 6.2] | 7.0 [3.5 to 12.1]
  Month 6: >=4 fold rise | 0.0 [0.0 to 6.7] | 9.2 [5.2 to 14.7] | 12.7 [7.9 to 18.9]
  Month 6: >=8 fold rise | 0.0 [0.0 to 6.7] | 6.1 [3.0 to 11.0] | 10.1 [5.9 to 15.9]
  Month 6: >=16 fold rise | 0.0 [0.0 to 6.7] | 1.2 [0.1 to 4.4] | 5.1 [2.2 to 9.7]
  Month 6: >=32 fold rise | 0.0 [0.0 to 6.7] | 0.6 [0.0 to 3.4] | 2.5 [0.7 to 6.4]
  Day 187: >=4 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=4 fold rise | 0.0 [0.0 to 6.7] | 63.0 [55.0 to 70.4] | 71.5 [63.8 to 78.4]
  Day 187: >=8 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=8 fold rise | 0.0 [0.0 to 6.7] | 43.8 [36.1 to 51.8] | 55.7 [47.6 to 63.6]
  Day 187: >=16 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=16 fold rise | 0.0 [0.0 to 6.7] | 16.7 [11.3 to 23.3] | 32.9 [25.7 to 40.8]
  Day 187: >=32 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=32 fold rise | 0.0 [0.0 to 6.7] | 5.6 [2.6 to 10.3] | 13.3 [8.4 to 19.6]
  Month 7: >=4 fold rise | 1.9 [0.0 to 10.1] | 91.4 [86.0 to 95.2] | 91.8 [86.3 to 95.5]
  Month 7: >=8 fold rise | 0.0 [0.0 to 6.7] | 76.7 [69.4 to 82.9] | 78.5 [71.2 to 84.6]
  Month 7: >=16 fold rise | 0.0 [0.0 to 6.7] | 47.2 [39.4 to 55.2] | 56.3 [48.2 to 64.2]
  Month 7: >=32 fold rise | 0.0 [0.0 to 6.7] | 20.2 [14.4 to 27.2] | 21.5 [15.4 to 28.8]
  Month 12: >=4 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=4 fold rise | 2.0 [0.0 to 10.4] | 50.6 [42.6 to 58.6] | 61.3 [53.1 to 69.0]
  Month 12: >=8 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=8 fold rise | 2.0 [0.0 to 10.4] | 27.5 [20.7 to 35.1] | 40.6 [32.8 to 48.8]
  Month 12: >=16 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=16 fold rise | 0.0 [0.0 to 7.0] | 9.4 [5.3 to 15.0] | 14.2 [9.1 to 20.7]
  Month 12: >=32 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=32 fold rise | 0.0 [0.0 to 7.0] | 2.5 [0.7 to 6.3] | 1.9 [0.4 to 5.6]
  Month 18: >=4 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=4 fold rise | 0.0 [0.0 to 7.0] | 27.9 [21.0 to 35.7] | 39.5 [31.6 to 47.7]
  Month 18: >=8 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=8 fold rise | 0.0 [0.0 to 7.0] | 13.6 [8.6 to 20.1] | 20.4 [14.3 to 27.7]
  Month 18: >=16 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=16 fold rise | 0.0 [0.0 to 7.0] | 5.8 [2.7 to 10.8] | 7.2 [3.7 to 12.6]
  Month 18: >=32 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=32 fold rise | 0.0 [0.0 to 7.0] | 1.3 [0.2 to 4.6] | 0.0 [0.0 to 2.4]

41. Secondary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Toxin B Specific Antibody Levels at Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Description: Toxin A antibodies were measured using neutralization assay.
Time Frame: Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants
  Day 30: >=4 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=4 fold rise | 3.8 [0.5 to 13.0] | 34.0 [26.7 to 41.8] | 43.3 [35.4 to 51.4]
  Day 30: >=8 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=8 fold rise | 1.9 [0.0 to 10.1] | 29.6 [22.7 to 37.3] | 38.9 [31.2 to 46.9]
  Day 30: >=16 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=16 fold rise | 1.9 [0.0 to 10.1] | 21.6 [15.5 to 28.7] | 30.6 [23.5 to 38.4]
  Day 30: >=32 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=32 fold rise | 0.0 [0.0 to 6.7] | 16.7 [11.3 to 23.3] | 20.4 [14.4 to 27.5]
  Day 37: >=4 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=4 fold rise | 3.8 [0.5 to 13.0] | 36.8 [29.4 to 44.7] | 47.8 [39.7 to 55.9]
  Day 37: >=8 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=8 fold rise | 1.9 [0.0 to 10.1] | 30.7 [23.7 to 38.4] | 42.7 [34.8 to 50.8]
  Day 37: >=16 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=16 fold rise | 1.9 [0.0 to 10.1] | 23.9 [17.6 to 31.2] | 33.1 [25.8 to 41.1]
  Day 37: >=32 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=32 fold rise | 0.0 [0.0 to 6.7] | 18.4 [12.8 to 25.2] | 22.3 [16.0 to 29.6]
  Month 2: >=4 fold rise | 3.8 [0.5 to 13.0] | 37.4 [30.0 to 45.3] | 47.5 [39.5 to 55.6]
  Month 2: >=8 fold rise | 1.9 [0.0 to 10.1] | 32.5 [25.4 to 40.3] | 39.9 [32.2 to 48.0]
  Month 2: >=16 fold rise | 1.9 [0.0 to 10.1] | 23.3 [17.1 to 30.6] | 29.7 [22.7 to 37.5]
  Month 2: >=32 fold rise | 1.9 [0.0 to 10.1] | 16.6 [11.2 to 23.2] | 23.4 [17.1 to 30.8]
  Month 6: >=4 fold rise | 3.8 [0.5 to 13.0] | 30.1 [23.1 to 37.7] | 41.1 [33.4 to 49.2]
  Month 6: >=8 fold rise | 3.8 [0.5 to 13.0] | 21.5 [15.4 to 28.6] | 32.3 [25.1 to 40.2]
  Month 6: >=16 fold rise | 1.9 [0.0 to 10.1] | 13.5 [8.7 to 19.7] | 21.5 [15.4 to 28.8]
  Month 6: >=32 fold rise | 0.0 [0.0 to 6.7] | 6.7 [3.4 to 11.8] | 12.0 [7.4 to 18.1]
  Day 187: >=4 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=4 fold rise | 1.9 [0.0 to 10.1] | 79.0 [71.9 to 85.0] | 87.3 [81.1 to 92.1]
  Day 187: >=8 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=8 fold rise | 1.9 [0.0 to 10.1] | 68.5 [60.8 to 75.6] | 78.5 [71.2 to 84.6]
  Day 187: >=16 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=16 fold rise | 1.9 [0.0 to 10.1] | 52.5 [44.5 to 60.4] | 63.3 [55.3 to 70.8]
  Day 187: >=32 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=32 fold rise | 0.0 [0.0 to 6.7] | 32.1 [25.0 to 39.9] | 46.2 [38.2 to 54.3]
  Month 7: >=4 fold rise | 3.8 [0.5 to 13.0] | 92.0 [86.7 to 95.7] | 93.7 [88.7 to 96.9]
  Month 7: >=8 fold rise | 1.9 [0.0 to 10.1] | 84.7 [78.2 to 89.8] | 90.5 [84.8 to 94.6]
  Month 7: >=16 fold rise | 1.9 [0.0 to 10.1] | 76.1 [68.8 to 82.4] | 83.5 [76.8 to 89.0]
  Month 7: >=32 fold rise | 1.9 [0.0 to 10.1] | 55.8 [47.9 to 63.6] | 66.5 [58.5 to 73.8]
  Month 12: >=4 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=4 fold rise | 3.9 [0.5 to 13.5] | 75.0 [67.6 to 81.5] | 85.8 [79.3 to 90.9]
  Month 12: >=8 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=8 fold rise | 3.9 [0.5 to 13.5] | 59.4 [51.3 to 67.1] | 73.5 [65.9 to 80.3]
  Month 12: >=16 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=16 fold rise | 3.9 [0.5 to 13.5] | 39.4 [31.8 to 47.4] | 51.6 [43.5 to 59.7]
  Month 12: >=32 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=32 fold rise | 0.0 [0.0 to 7.0] | 18.1 [12.5 to 25.0] | 27.1 [20.3 to 34.8]
  Month 18: >=4 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=4 fold rise | 7.8 [2.2 to 18.9] | 66.9 [58.9 to 74.2] | 78.3 [70.9 to 84.6]
  Month 18: >=8 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=8 fold rise | 3.9 [0.5 to 13.5] | 44.2 [36.2 to 52.4] | 60.5 [52.3 to 68.4]
  Month 18: >=16 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=16 fold rise | 2.0 [0.0 to 10.4] | 29.2 [22.2 to 37.1] | 40.1 [32.3 to 48.4]
  Month 18: >=32 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=32 fold rise | 0.0 [0.0 to 7.0] | 13.0 [8.1 to 19.3] | 23.0 [16.6 to 30.5]

42. Secondary Outcome: Month 0, 1 and 6 Regimen: Percentage of Participants Achieving>=4,>=8,>=16,>=32 Fold Rise From Baseline in Both Toxin A and Toxin B Antibody Levels at Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Description: Toxin A and toxin B antibodies were measured using neutralization assay.
Time Frame: Day 30, 37, 187 and Month 2, 6, 7, 12, 18
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo: Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(100 mcg):Month0, 1and 6 Regimen | Clostridium Difficile Vaccine(200 mcg):Month0, 1and 6 Regimen
Number analyzed (Participants) | 53 | 163 | 158
percentage of participants
  Day 30: >=4 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=4 fold rise | 0.0 [0.0 to 6.7] | 11.7 [7.2 to 17.7] | 12.1 [7.4 to 18.3]
  Day 30: >=8 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=8 fold rise | 0.0 [0.0 to 6.7] | 9.3 [5.3 to 14.8] | 9.6 [5.4 to 15.3]
  Day 30: >=16 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=16 fold rise | 0.0 [0.0 to 6.7] | 3.1 [1.0 to 7.1] | 7.0 [3.5 to 12.2]
  Day 30: >=32 fold rise: number analyzed (Participants) | 53 | 162 | 157
  Day 30: >=32 fold rise | 0.0 [0.0 to 6.7] | 0.6 [0.0 to 3.4] | 3.2 [1.0 to 7.3]
  Day 37: >=4 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=4 fold rise | 0.0 [0.0 to 6.7] | 19.0 [13.3 to 25.9] | 26.8 [20.0 to 34.4]
  Day 37: >=8 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=8 fold rise | 0.0 [0.0 to 6.7] | 9.2 [5.2 to 14.7] | 19.7 [13.8 to 26.8]
  Day 37: >=16 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=16 fold rise | 0.0 [0.0 to 6.7] | 3.7 [1.4 to 7.8] | 8.3 [4.5 to 13.7]
  Day 37: >=32 fold rise: number analyzed (Participants) | 53 | 163 | 157
  Day 37: >=32 fold rise | 0.0 [0.0 to 6.7] | 1.2 [0.1 to 4.4] | 3.8 [1.4 to 8.1]
  Month 2: >=4 fold rise | 1.9 [0.0 to 10.1] | 18.4 [12.8 to 25.2] | 24.1 [17.6 to 31.5]
  Month 2: >=8 fold rise | 0.0 [0.0 to 6.7] | 10.4 [6.2 to 16.2] | 14.6 [9.5 to 21.0]
  Month 2: >=16 fold rise | 0.0 [0.0 to 6.7] | 3.1 [1.0 to 7.0] | 7.0 [3.5 to 12.1]
  Month 2: >=32 fold rise | 0.0 [0.0 to 6.7] | 1.2 [0.1 to 4.4] | 3.2 [1.0 to 7.2]
  Month 6: >=4 fold rise | 0.0 [0.0 to 6.7] | 8.0 [4.3 to 13.3] | 10.1 [5.9 to 15.9]
  Month 6: >=8 fold rise | 0.0 [0.0 to 6.7] | 2.5 [0.7 to 6.2] | 6.3 [3.1 to 11.3]
  Month 6: >=16 fold rise | 0.0 [0.0 to 6.7] | 0.6 [0.0 to 3.4] | 2.5 [0.7 to 6.4]
  Month 6: >=32 fold rise | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 2.2] | 1.3 [0.2 to 4.5]
  Day 187: >=4 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=4 fold rise | 0.0 [0.0 to 6.7] | 58.6 [50.6 to 66.3] | 69.6 [61.8 to 76.7]
  Day 187: >=8 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=8 fold rise | 0.0 [0.0 to 6.7] | 39.5 [31.9 to 47.5] | 50.6 [42.6 to 58.7]
  Day 187: >=16 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=16 fold rise | 0.0 [0.0 to 6.7] | 11.1 [6.7 to 17.0] | 27.2 [20.4 to 34.9]
  Day 187: >=32 fold rise: number analyzed (Participants) | 53 | 162 | 158
  Day 187: >=32 fold rise | 0.0 [0.0 to 6.7] | 2.5 [0.7 to 6.2] | 10.8 [6.4 to 16.7]
  Month 7: >=4 fold rise | 0.0 [0.0 to 6.7] | 84.7 [78.2 to 89.8] | 87.3 [81.1 to 92.1]
  Month 7: >=8 fold rise | 0.0 [0.0 to 6.7] | 68.7 [61.0 to 75.7] | 74.1 [66.5 to 80.7]
  Month 7: >=16 fold rise | 0.0 [0.0 to 6.7] | 41.1 [33.5 to 49.1] | 52.5 [44.4 to 60.5]
  Month 7: >=32 fold rise | 0.0 [0.0 to 6.7] | 14.1 [9.2 to 20.4] | 17.1 [11.6 to 23.9]
  Month 12: >=4 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=4 fold rise | 0.0 [0.0 to 7.0] | 44.4 [36.5 to 52.4] | 58.7 [50.5 to 66.5]
  Month 12: >=8 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=8 fold rise | 0.0 [0.0 to 7.0] | 21.9 [15.7 to 29.1] | 35.5 [28.0 to 43.6]
  Month 12: >=16 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=16 fold rise | 0.0 [0.0 to 7.0] | 5.0 [2.2 to 9.6] | 9.7 [5.5 to 15.5]
  Month 12: >=32 fold rise: number analyzed (Participants) | 51 | 160 | 155
  Month 12: >=32 fold rise | 0.0 [0.0 to 7.0] | 1.3 [0.2 to 4.4] | 1.3 [0.2 to 4.6]
  Month 18: >=4 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=4 fold rise | 0.0 [0.0 to 7.0] | 23.4 [16.9 to 30.9] | 36.2 [28.6 to 44.4]
  Month 18: >=8 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=8 fold rise | 0.0 [0.0 to 7.0] | 10.4 [6.1 to 16.3] | 19.1 [13.2 to 26.2]
  Month 18: >=16 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=16 fold rise | 0.0 [0.0 to 7.0] | 3.9 [1.4 to 8.3] | 3.9 [1.5 to 8.4]
  Month 18: >=32 fold rise: number analyzed (Participants) | 51 | 154 | 152
  Month 18: >=32 fold rise | 0.0 [0.0 to 7.0] | 0.6 [0.0 to 3.6] | 0.0 [0.0 to 2.4]

43. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin A at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin A antibodies (threshold >= 219 neutralization units/mL) were measured using neutralization assay.
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: Evaluable immunogenicity population: All eligible participants re-randomized to the extension stage of study, who received fourth study vaccination with formulation to which they were randomized, had at least 1 valid assay result from blood drawn within 7 to 14 days after Vaccination 4 and had no major protocol violations. Here, 'Number Analyzed' signifies participants evaluable for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 100 mcg dose level received a fourth dose of Clostridium difficile vaccine intramuscularly at the 100 mcg dose level in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
percentage of participants
  Day 1 | 6.3 [0.2 to 30.2] | 22.2 [6.4 to 47.6] | 20.8 [7.1 to 42.2] | 30.0 [11.9 to 54.3]
  Day 8 | 6.3 [0.2 to 30.2] | 100.0 [81.5 to 100.0] | 12.5 [2.7 to 32.4] | 100.0 [83.2 to 100.0]
  Day 30 | 6.3 [0.2 to 30.2] | 100.0 [81.5 to 100.0] | 29.2 [12.6 to 51.1] | 100.0 [83.2 to 100.0]
  Month 6: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6 | 6.3 [0.2 to 30.2] | 100.0 [81.5 to 100.0] | 21.7 [7.5 to 43.7] | 100.0 [83.2 to 100.0]
  Month 12: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12 | 6.3 [0.2 to 30.2] | 88.9 [65.3 to 98.6] | 14.3 [3.0 to 36.3] | 95.0 [75.1 to 99.9]
  Month 18: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18 | 12.5 [1.6 to 38.3] | 82.4 [56.6 to 96.2] | 15.0 [3.2 to 37.9] | 95.0 [75.1 to 99.9]
  Month 24: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24 | 6.3 [0.2 to 30.2] | 82.4 [56.6 to 96.2] | 5.0 [0.1 to 24.9] | 84.2 [60.4 to 96.6]
  Month 30: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30 | 7.1 [0.2 to 33.9] | 76.5 [50.1 to 93.2] | 10.0 [1.2 to 31.7] | 94.4 [72.7 to 99.9]
  Month 36: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36 | 7.7 [0.2 to 36.0] | 87.5 [61.7 to 98.4] | 10.0 [1.2 to 31.7] | 94.4 [72.7 to 99.9]

44. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin B at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin B antibodies (threshold >= 2586 neutralization units/mL) were measured using neutralization assay.
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
percentage of participants
  Day 1 | 12.5 [1.6 to 38.3] | 44.4 [21.5 to 69.2] | 29.2 [12.6 to 51.1] | 40.0 [19.1 to 63.9]
  Day 8 | 12.5 [1.6 to 38.3] | 88.9 [65.3 to 98.6] | 25.0 [9.8 to 46.7] | 95.0 [75.1 to 99.9]
  Day 30 | 12.5 [1.6 to 38.3] | 100.0 [81.5 to 100.0] | 25.0 [9.8 to 46.7] | 95.0 [75.1 to 99.9]
  Month 6: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6 | 6.3 [0.2 to 30.2] | 94.4 [72.7 to 99.9] | 21.7 [7.5 to 43.7] | 85.0 [62.1 to 96.8]
  Month 12: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12 | 6.3 [0.2 to 30.2] | 88.9 [65.3 to 98.6] | 19.0 [5.4 to 41.9] | 85.0 [62.1 to 96.8]
  Month 18: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18 | 0.0 [0.0 to 20.6] | 82.4 [56.6 to 96.2] | 30.0 [11.9 to 54.3] | 75.0 [50.9 to 91.3]
  Month 24: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24 | 0.0 [0.0 to 20.6] | 64.7 [38.3 to 85.8] | 25.0 [8.7 to 49.1] | 78.9 [54.4 to 93.9]
  Month 30: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30 | 0.0 [0.0 to 23.2] | 70.6 [44.0 to 89.7] | 25.0 [8.7 to 49.1] | 77.8 [52.4 to 93.6]
  Month 36: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36 | 0.0 [0.0 to 24.7] | 75.0 [47.6 to 92.7] | 25.0 [8.7 to 49.1] | 77.8 [52.4 to 93.6]

45. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Both Toxin A and Toxin B at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin A and B antibodies (threshold >= 219 and 2586 neutralization units/mL) were measured using neutralization assay.
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
percentage of participants
  Day 1 | 0.0 [0.0 to 20.6] | 11.1 [1.4 to 34.7] | 8.3 [1.0 to 27.0] | 15.0 [3.2 to 37.9]
  Day 8 | 0.0 [0.0 to 20.6] | 88.9 [65.3 to 98.6] | 4.2 [0.1 to 21.1] | 95.0 [75.1 to 99.9]
  Day 30 | 0.0 [0.0 to 20.6] | 100.0 [81.5 to 100.0] | 8.3 [1.0 to 27.0] | 95.0 [75.1 to 99.9]
  Month 6: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6 | 0.0 [0.0 to 20.6] | 94.4 [72.7 to 99.9] | 8.7 [1.1 to 28.0] | 85.0 [62.1 to 96.8]
  Month 12: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12 | 0.0 [0.0 to 20.6] | 83.3 [58.6 to 96.4] | 9.5 [1.2 to 30.4] | 80.0 [56.3 to 94.3]
  Month 18: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18 | 0.0 [0.0 to 20.6] | 70.6 [44.0 to 89.7] | 10.0 [1.2 to 31.7] | 75.0 [50.9 to 91.3]
  Month 24: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24 | 0.0 [0.0 to 20.6] | 52.9 [27.8 to 77.0] | 0.0 [0.0 to 16.8] | 73.7 [48.8 to 90.9]
  Month 30: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30 | 0.0 [0.0 to 23.2] | 58.8 [32.9 to 81.6] | 10.0 [1.2 to 31.7] | 72.2 [46.5 to 90.3]
  Month 36: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36 | 0.0 [0.0 to 24.7] | 68.8 [41.3 to 89.0] | 10.0 [1.2 to 31.7] | 77.8 [52.4 to 93.6]

46. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin A at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin A antibodies (threshold >= 219 neutralization units/mL) were measured using neutralization assay.
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 100 mcg dose level received fourth dose of Clostridium difficile vaccine intramuscularly at the 100 mcg dose level in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
- 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 200 mcg dose level received placebo as the fourth dose in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
percentage of participants
  Day 1 | 54.2 [39.2 to 68.6] | 32.7 [20.3 to 47.1] | 50.0 [36.6 to 63.4] | 61.0 [47.4 to 73.5]
  Day 8 | 50.0 [35.2 to 64.8] | 94.2 [84.1 to 98.8] | 53.4 [39.9 to 66.7] | 94.9 [85.9 to 98.9]
  Day 30 | 37.5 [24.0 to 52.6] | 100.0 [93.2 to 100.0] | 56.9 [43.2 to 69.8] | 100.0 [93.9 to 100.0]
  Month 6: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6 | 40.4 [26.4 to 55.7] | 98.0 [89.4 to 99.9] | 47.4 [34.0 to 61.0] | 96.6 [88.3 to 99.6]
  Month 12: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12 | 34.8 [21.4 to 50.2] | 88.0 [75.7 to 95.5] | 47.3 [33.7 to 61.2] | 96.6 [88.1 to 99.6]
  Month 18: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18 | 20.5 [9.8 to 35.3] | 73.5 [58.9 to 85.1] | 25.9 [15.0 to 39.7] | 91.4 [81.0 to 97.1]
  Month 24: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24 | 38.6 [24.4 to 54.5] | 68.8 [53.7 to 81.3] | 37.7 [24.8 to 52.1] | 77.2 [64.2 to 87.3]
  Month 30: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30 | 19.5 [8.8 to 34.9] | 60.0 [44.3 to 74.3] | 29.4 [17.5 to 43.8] | 72.7 [59.0 to 83.9]
  Month 36: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36 | 22.0 [10.6 to 37.6] | 45.5 [30.4 to 61.2] | 24.0 [13.1 to 38.2] | 71.7 [57.7 to 83.2]

47. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Toxin B at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin B antibodies (threshold >= 2586 neutralization units/mL) were measured using neutralization assay.
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
percentage of participants
  Day 1 | 39.6 [25.8 to 54.7] | 15.4 [6.9 to 28.1] | 41.4 [28.6 to 55.1] | 50.8 [37.5 to 64.1]
  Day 8 | 33.3 [20.4 to 48.4] | 69.2 [54.9 to 81.3] | 36.2 [24.0 to 49.9] | 91.5 [81.3 to 97.2]
  Day 30 | 35.4 [22.2 to 50.5] | 86.5 [74.2 to 94.4] | 43.1 [30.2 to 56.8] | 96.6 [88.3 to 99.6]
  Month 6: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6 | 31.9 [19.1 to 47.1] | 70.0 [55.4 to 82.1] | 47.4 [34.0 to 61.0] | 86.4 [75.0 to 94.0]
  Month 12: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12 | 32.6 [19.5 to 48.0] | 62.0 [47.2 to 75.3] | 43.6 [30.3 to 57.7] | 82.8 [70.6 to 91.4]
  Month 18: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18 | 27.3 [15.0 to 42.8] | 42.9 [28.8 to 57.8] | 35.2 [22.7 to 49.4] | 55.2 [41.5 to 68.3]
  Month 24: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24 | 50.0 [34.6 to 65.4] | 31.3 [18.7 to 46.3] | 35.8 [23.1 to 50.2] | 52.6 [39.0 to 66.0]
  Month 30: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30 | 31.7 [18.1 to 48.1] | 31.1 [18.2 to 46.6] | 29.4 [17.5 to 43.8] | 58.2 [44.1 to 71.3]
  Month 36: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36 | 29.3 [16.1 to 45.5] | 27.3 [15.0 to 42.8] | 26.0 [14.6 to 40.3] | 52.8 [38.6 to 66.7]

48. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Percentage of Participants Achieving Prespecified Antibody Titer Level for Both Toxin A and Toxin B at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin A and B antibodies (threshold >= 219 and 2586 neutralization units/mL) were measured using neutralization assay.
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
percentage of participants
  Day 1 | 29.2 [17.0 to 44.1] | 9.6 [3.2 to 21.0] | 27.6 [16.7 to 40.9] | 40.7 [28.1 to 54.3]
  Day 8 | 25.0 [13.6 to 39.6] | 69.2 [54.9 to 81.3] | 25.9 [15.3 to 39.0] | 89.8 [79.2 to 96.2]
  Day 30 | 25.0 [13.6 to 39.6] | 86.5 [74.2 to 94.4] | 29.3 [18.1 to 42.7] | 96.6 [88.3 to 99.6]
  Month 6: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6 | 19.1 [9.1 to 33.3] | 70.0 [55.4 to 82.1] | 29.8 [18.4 to 43.4] | 84.7 [73.0 to 92.8]
  Month 12: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12 | 17.4 [7.8 to 31.4] | 62.0 [47.2 to 75.3] | 25.5 [14.7 to 39.0] | 81.0 [68.6 to 90.1]
  Month 18: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18 | 9.1 [2.5 to 21.7] | 40.8 [27.0 to 55.8] | 14.8 [6.6 to 27.1] | 53.4 [39.9 to 66.7]
  Month 24: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24 | 22.7 [11.5 to 37.8] | 29.2 [17.0 to 44.1] | 26.4 [15.3 to 40.3] | 50.9 [37.3 to 64.4]
  Month 30: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30 | 12.2 [4.1 to 26.2] | 22.2 [11.2 to 37.1] | 15.7 [7.0 to 28.6] | 47.3 [33.7 to 61.2]
  Month 36: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36 | 9.8 [2.7 to 23.1] | 18.2 [8.2 to 32.7] | 8.0 [2.2 to 19.2] | 45.3 [31.6 to 59.6]

49. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Geometric Mean Concentration for Toxin A Specific Neutralizing Antibody Levels at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: as for outcome 31
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: neutralization units per milliliter
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
neutralization units per milliliter
  Day 1 | 88 [70.1 to 110.1] | 142 [90.7 to 221.6] | 120 [90.9 to 159.2] | 198 [111.4 to 351.8]
  Day 8 | 88 [74.9 to 103.6] | 2161 [1199.3 to 3895.6] | 118 [92.1 to 149.9] | 3787 [1885.2 to 7608.4]
  Day 30 | 95 [70.4 to 128.3] | 5446 [3389.1 to 8751.2] | 126 [95.3 to 165.5] | 8013 [5104.5 to 12578.9]
  Month 6: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6 | 89 [69.0 to 114.9] | 1745 [1061.2 to 2870.5] | 109 [84.7 to 140.3] | 2686 [1640.9 to 4397.2]
  Month 12: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12 | 87 [70.4 to 108.6] | 908 [602.7 to 1367.0] | 96 [76.6 to 120.6] | 1417 [892.5 to 2249.6]
  Month 18: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18 | 96 [71.7 to 128.3] | 666 [393.0 to 1129.3] | 102 [78.7 to 131.8] | 925 [623.8 to 1372.1]
  Month 24: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24 | 85 [72.9 to 98.5] | 447 [276.9 to 722.8] | 95 [79.5 to 113.0] | 659 [399.6 to 1087.2]
  Month 30: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30 | 87 [70.9 to 106.1] | 468 [291.8 to 749.7] | 92 [77.1 to 110.1] | 656 [448.0 to 961.7]
  Month 36: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36 | 89 [68.2 to 117.5] | 495 [294.3 to 832.1] | 96 [79.3 to 116.0] | 774 [492.1 to 1216.6]

50. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Geometric Mean Concentration for Toxin B Specific Neutralizing Antibody Levels at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: as for outcome 30
Time Frame: Extension Stage Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: neutralization units per milliliter
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
neutralization units per milliliter
  Day 1 | 267 [135.4 to 524.8] | 1352 [637.0 to 2871.7] | 791 [348.6 to 1792.5] | 1632 [626.0 to 4256.6]
  Day 8 | 256 [135.7 to 482.0] | 14754 [6929.5 to 31414.7] | 807 [331.2 to 1968.2] | 18832 [8516.0 to 41644.3]
  Day 30 | 289 [149.7 to 559.0] | 25297 [15053.2 to 42513.1] | 939 [406.4 to 2169.6] | 50637 [26616.8 to 96335.4]
  Month 6: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6 | 322 [169.2 to 613.1] | 12467 [7673.0 to 20257.7] | 876 [356.0 to 2154.5] | 19239 [9155.7 to 40426.7]
  Month 12: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12 | 298 [162.3 to 545.2] | 6707 [4294.7 to 10475.5] | 787 [308.1 to 2009.2] | 11126 [5350.8 to 23136.3]
  Month 18: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18 | 216 [127.4 to 365.6] | 5428 [3375.7 to 8728.5] | 941 [342.2 to 2587.5] | 8340 [3977.0 to 17489.0]
  Month 24: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24 | 211 [125.1 to 355.6] | 3530 [2312.5 to 5387.9] | 932 [360.3 to 2408.7] | 7101 [3501.0 to 14403.0]
  Month 30: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30 | 221 [122.6 to 399.0] | 3373 [2150.1 to 5290.8] | 709 [273.2 to 1841.3] | 6061 [3387.3 to 10846.4]
  Month 36: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36 | 239 [113.2 to 505.4] | 3457 [2137.7 to 5590.4] | 689 [280.2 to 1694.7] | 7115 [3694.4 to 13701.5]

51. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Geometric Mean Concentration for Toxin A Specific Neutralizing Antibody Levels at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: as for outcome 31
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: neutralization units per milliliter
Groups:
- 100mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen: Eligible participants who received the first 3 doses of Clostridium difficile vaccine at the 100 mcg dose level received placebo intramuscularly as the fourth dose in extension stage at visit 9 (340 to 380 Days after vaccination 3). Participants were followed up to 36 months after the last vaccination.
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
neutralization units per milliliter
  Day 1 | 230 [173.7 to 304.7] | 152 [120.7 to 192.4] | 249 [185.3 to 334.0] | 281 [212.4 to 372.9]
  Day 8 | 235 [182.2 to 303.6] | 1188 [880.5 to 1603.8] | 271 [202.0 to 362.6] | 2300 [1709.2 to 3095.2]
  Day 30 | 200 [151.8 to 264.0] | 3288 [2464.9 to 4384.7] | 283 [211.8 to 376.9] | 4695 [3469.1 to 6352.8]
  Month 6: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6 | 172 [129.3 to 227.7] | 1107 [864.9 to 1415.8] | 227 [167.3 to 307.0] | 1538 [1195.0 to 1980.3]
  Month 12: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12 | 163 [118.8 to 223.2] | 649 [502.8 to 838.5] | 211 [159.6 to 280.2] | 982 [802.8 to 1201.6]
  Month 18: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18 | 130 [99.5 to 170.9] | 348 [266.1 to 456.2] | 139 [107.7 to 180.4] | 497 [395.3 to 624.8]
  Month 24: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24 | 173 [130.9 to 229.8] | 298 [227.3 to 391.5] | 193 [147.3 to 254.1] | 438 [337.6 to 569.2]
  Month 30: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30 | 120 [94.2 to 153.5] | 273 [216.3 to 343.5] | 146 [115.0 to 185.5] | 386 [295.3 to 505.3]
  Month 36: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36 | 129 [99.1 to 168.5] | 222 [174.0 to 284.0] | 141 [111.2 to 179.5] | 355 [276.6 to 455.8]

52. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Geometric Mean Concentration for Toxin B Specific Neutralizing Antibody Levels at Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: as for outcome 30
Time Frame: Days 1, 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: neutralization units per milliliter
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
neutralization units per milliliter
  Day 1 | 1424 [891.9 to 2273.8] | 704 [480.8 to 1031.1] | 1925 [1220.4 to 3037.8] | 2186 [1483.4 to 3220.4]
  Day 8 | 1347 [823.7 to 2201.9] | 5011 [3346.2 to 7504.7] | 1862 [1179.8 to 2938.7] | 17205 [12065.9 to 24534.4]
  Day 30 | 1328 [819.3 to 2151.5] | 11885 [7950.3 to 17768.1] | 1776 [1185.2 to 2661.8] | 32905 [23885.1 to 45330.7]
  Month 6: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6 | 1258 [789.4 to 2004.7] | 4306 [2991.0 to 6200.4] | 2056 [1315.2 to 3212.9] | 10842 [7872.3 to 14930.8]
  Month 12: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12 | 1207 [735.7 to 1979.2] | 2693 [1856.1 to 3906.0] | 1681 [1102.4 to 2563.7] | 7126 [5159.1 to 9843.7]
  Month 18: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18 | 875 [550.5 to 1389.7] | 1587 [1033.5 to 2437.7] | 997 [639.4 to 1555.0] | 3079 [2254.0 to 4205.8]
  Month 24: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24 | 1613 [983.7 to 2643.9] | 1464 [925.8 to 2313.9] | 1436 [900.1 to 2289.6] | 3299 [2323.1 to 4684.7]
  Month 30: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30 | 911 [548.4 to 1513.6] | 1400 [945.9 to 2072.9] | 1227 [831.6 to 1809.0] | 3027 [2179.6 to 4204.5]
  Month 36: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36 | 885 [523.8 to 1494.8] | 1165 [751.0 to 1808.4] | 1021 [689.4 to 1511.1] | 2408 [1785.1 to 3247.1]

53. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Geometric Mean Fold Rise in Toxin A Specific Neutralizing Antibody Levels From Baseline at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: as for outcome 35
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
fold rise
  Day 8 | 1.00 [0.88 to 1.15] | 15.25 [8.57 to 27.11] | 0.98 [0.84 to 1.14] | 19.13 [9.09 to 40.28]
  Day 30 | 1.08 [0.96 to 1.22] | 38.41 [21.07 to 70.02] | 1.04 [0.87 to 1.26] | 40.47 [18.52 to 88.48]
  Month 6: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6 | 1.01 [0.98 to 1.04] | 12.31 [6.45 to 23.51] | 0.95 [0.77 to 1.17] | 13.57 [7.33 to 25.10]
  Month 12: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12 | 1.00 [0.99 to 1.00] | 6.40 [3.55 to 11.55] | 0.90 [0.71 to 1.15] | 7.16 [3.95 to 12.98]
  Month 18: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18 | 1.09 [0.84 to 1.42] | 4.54 [2.47 to 8.33] | 0.94 [0.73 to 1.22] | 4.67 [2.61 to 8.37]
  Month 24: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24 | 0.97 [0.73 to 1.28] | 3.05 [1.81 to 5.14] | 0.88 [0.68 to 1.14] | 3.29 [1.71 to 6.34]
  Month 30: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30 | 0.97 [0.92 to 1.03] | 3.19 [1.89 to 5.39] | 0.85 [0.67 to 1.09] | 3.32 [1.94 to 5.67]
  Month 36: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36 | 0.99 [0.98 to 1.01] | 3.74 [2.32 to 6.03] | 0.89 [0.72 to 1.10] | 3.91 [2.09 to 7.33]

54. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Geometric Mean Fold Rise in Toxin B Specific Neutralizing Antibody Levels From Baseline at Day 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: as for outcome 34
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
fold rise
  Day 8 | 0.96 [0.78 to 1.18] | 10.91 [6.02 to 19.75] | 1.02 [0.84 to 1.25] | 11.54 [5.70 to 23.34]
  Day 30 | 1.09 [0.90 to 1.30] | 18.70 [9.46 to 36.99] | 1.19 [1.03 to 1.36] | 31.02 [13.73 to 70.07]
  Month 6: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6 | 1.21 [0.94 to 1.55] | 9.22 [4.62 to 18.39] | 1.09 [0.90 to 1.31] | 11.79 [5.68 to 24.44]
  Month 12: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12 | 1.12 [0.79 to 1.58] | 4.96 [2.76 to 8.91] | 0.93 [0.76 to 1.15] | 6.82 [3.39 to 13.69]
  Month 18: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18 | 0.81 [0.58 to 1.13] | 3.49 [1.96 to 6.22] | 1.02 [0.75 to 1.38] | 5.11 [2.28 to 11.44]
  Month 24: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24 | 0.79 [0.50 to 1.26] | 2.27 [1.26 to 4.09] | 1.01 [0.72 to 1.41] | 3.80 [1.88 to 7.66]
  Month 30: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30 | 0.74 [0.50 to 1.11] | 2.17 [1.30 to 3.61] | 0.77 [0.58 to 1.00] | 3.13 [1.41 to 6.96]
  Month 36: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36 | 0.87 [0.65 to 1.16] | 2.40 [1.52 to 3.79] | 0.74 [0.57 to 0.98] | 3.68 [1.78 to 7.59]

55. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Geometric Mean Fold Rise in Toxin A Specific Neutralizing Antibody Levels From Baseline at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: as for outcome 35
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
fold rise
  Day 8 | 1.02 [0.90 to 1.16] | 7.80 [5.74 to 10.59] | 1.09 [0.97 to 1.22] | 8.17 [5.97 to 11.19]
  Day 30 | 0.87 [0.76 to 1.00] | 21.57 [16.24 to 28.65] | 1.14 [1.01 to 1.28] | 16.68 [11.72 to 23.74]
  Month 6: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6 | 0.74 [0.67 to 0.83] | 7.07 [5.22 to 9.58] | 0.89 [0.76 to 1.05] | 5.47 [4.19 to 7.13]
  Month 12: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12 | 0.71 [0.60 to 0.83] | 4.15 [3.10 to 5.55] | 0.85 [0.74 to 0.98] | 3.41 [2.69 to 4.34]
  Month 18: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18 | 0.57 [0.46 to 0.72] | 2.24 [1.65 to 3.04] | 0.55 [0.46 to 0.65] | 1.73 [1.36 to 2.20]
  Month 24: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24 | 0.76 [0.56 to 1.04] | 1.89 [1.40 to 2.55] | 0.75 [0.57 to 1.00] | 1.55 [1.17 to 2.03]
  Month 30: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30 | 0.51 [0.42 to 0.62] | 1.76 [1.33 to 2.34] | 0.56 [0.47 to 0.67] | 1.34 [1.03 to 1.74]
  Month 36: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36 | 0.55 [0.43 to 0.70] | 1.45 [1.03 to 2.03] | 0.53 [0.43 to 0.66] | 1.22 [0.91 to 1.64]

56. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Geometric Mean Fold Rise in Toxin B Specific Neutralizing Antibody Levels From Baseline at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: as for outcome 34
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
fold rise
  Day 8 | 0.95 [0.82 to 1.09] | 7.12 [4.98 to 10.16] | 0.97 [0.88 to 1.07] | 7.87 [5.60 to 11.06]
  Day 30 | 0.93 [0.81 to 1.07] | 16.88 [11.25 to 25.33] | 0.92 [0.79 to 1.07] | 15.05 [10.49 to 21.60]
  Month 6: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6 | 0.86 [0.77 to 0.95] | 5.97 [4.22 to 8.45] | 1.08 [0.86 to 1.36] | 4.96 [3.79 to 6.49]
  Month 12: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12 | 0.81 [0.69 to 0.95] | 3.73 [2.69 to 5.17] | 0.89 [0.71 to 1.11] | 3.10 [2.47 to 3.89]
  Month 18: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18 | 0.58 [0.42 to 0.79] | 2.25 [1.49 to 3.38] | 0.51 [0.40 to 0.65] | 1.34 [1.06 to 1.70]
  Month 24: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24 | 1.07 [0.61 to 1.86] | 2.00 [1.19 to 3.34] | 0.70 [0.50 to 0.98] | 1.45 [1.09 to 1.93]
  Month 30: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30 | 0.58 [0.41 to 0.80] | 2.09 [1.40 to 3.13] | 0.60 [0.47 to 0.77] | 1.36 [1.00 to 1.84]
  Month 36: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36 | 0.56 [0.35 to 0.89] | 1.85 [1.23 to 2.78] | 0.47 [0.37 to 0.61] | 1.09 [0.82 to 1.44]

57. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Toxin A Specific Antibody Levels at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin A antibodies were measured using neutralization assay.
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 20.6] | 88.9 [65.3 to 98.6] | 0.0 [0.0 to 14.2] | 85.0 [62.1 to 96.8]
  Day 8: >=8 fold rise | 0.0 [0.0 to 20.6] | 66.7 [41.0 to 86.7] | 0.0 [0.0 to 14.2] | 70.0 [45.7 to 88.1]
  Day 8: >=16 fold rise | 0.0 [0.0 to 20.6] | 38.9 [17.3 to 64.3] | 0.0 [0.0 to 14.2] | 70.0 [45.7 to 88.1]
  Day 8: >=32 fold rise | 0.0 [0.0 to 20.6] | 33.3 [13.3 to 59.0] | 0.0 [0.0 to 14.2] | 35.0 [15.4 to 59.2]
  Day 30: >=4 fold rise | 0.0 [0.0 to 20.6] | 100.0 [81.5 to 100.0] | 0.0 [0.0 to 14.2] | 90.0 [68.3 to 98.8]
  Day 30: >=8 fold rise | 0.0 [0.0 to 20.6] | 88.9 [65.3 to 98.6] | 0.0 [0.0 to 14.2] | 85.0 [62.1 to 96.8]
  Day 30: >=16 fold rise | 0.0 [0.0 to 20.6] | 72.2 [46.5 to 90.3] | 0.0 [0.0 to 14.2] | 75.0 [50.9 to 91.3]
  Day 30: >=32 fold rise | 0.0 [0.0 to 20.6] | 50.0 [26.0 to 74.0] | 0.0 [0.0 to 14.2] | 55.0 [31.5 to 76.9]
  Month 6: >=4 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=4 fold rise | 0.0 [0.0 to 20.6] | 72.2 [46.5 to 90.3] | 0.0 [0.0 to 14.8] | 80.0 [56.3 to 94.3]
  Month 6: >=8 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=8 fold rise | 0.0 [0.0 to 20.6] | 61.1 [35.7 to 82.7] | 0.0 [0.0 to 14.8] | 75.0 [50.9 to 91.3]
  Month 6: >=16 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=16 fold rise | 0.0 [0.0 to 20.6] | 44.4 [21.5 to 69.2] | 0.0 [0.0 to 14.8] | 40.0 [19.1 to 63.9]
  Month 6: >=32 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=32 fold rise | 0.0 [0.0 to 20.6] | 16.7 [3.6 to 41.4] | 0.0 [0.0 to 14.8] | 25.0 [8.7 to 49.1]
  Month 12: >=4 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=4 fold rise | 0.0 [0.0 to 20.6] | 72.2 [46.5 to 90.3] | 4.8 [0.1 to 23.8] | 65.0 [40.8 to 84.6]
  Month 12: >=8 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=8 fold rise | 0.0 [0.0 to 20.6] | 50.0 [26.0 to 74.0] | 0.0 [0.0 to 16.1] | 50.0 [27.2 to 72.8]
  Month 12: >=16 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=16 fold rise | 0.0 [0.0 to 20.6] | 27.8 [9.7 to 53.5] | 0.0 [0.0 to 16.1] | 30.0 [11.9 to 54.3]
  Month 12: >=32 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=32 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 16.1] | 5.0 [0.1 to 24.9]
  Month 18: >=4 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=4 fold rise | 6.3 [0.2 to 30.2] | 47.1 [23.0 to 72.2] | 0.0 [0.0 to 16.8] | 55.0 [31.5 to 76.9]
  Month 18: >=8 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=8 fold rise | 0.0 [0.0 to 20.6] | 41.2 [18.4 to 67.1] | 0.0 [0.0 to 16.8] | 45.0 [23.1 to 68.5]
  Month 18: >=16 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=16 fold rise | 0.0 [0.0 to 20.6] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 16.8] | 15.0 [3.2 to 37.9]
  Month 18: >=32 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=32 fold rise | 0.0 [0.0 to 20.6] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 16.8] | 5.0 [0.1 to 24.9]
  Month 24: >=4 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=4 fold rise | 0.0 [0.0 to 20.6] | 41.2 [18.4 to 67.1] | 0.0 [0.0 to 16.8] | 47.4 [24.4 to 71.1]
  Month 24: >=8 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=8 fold rise | 0.0 [0.0 to 20.6] | 23.5 [6.8 to 49.9] | 0.0 [0.0 to 16.8] | 31.6 [12.6 to 56.6]
  Month 24: >=16 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=16 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 15.8 [3.4 to 39.6]
  Month 24: >=32 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=32 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 5.3 [0.1 to 26.0]
  Month 30: >=4 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=4 fold rise | 0.0 [0.0 to 23.2] | 29.4 [10.3 to 56.0] | 0.0 [0.0 to 16.8] | 38.9 [17.3 to 64.3]
  Month 30: >=8 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=8 fold rise | 0.0 [0.0 to 23.2] | 17.6 [3.8 to 43.4] | 0.0 [0.0 to 16.8] | 16.7 [3.6 to 41.4]
  Month 30: >=16 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=16 fold rise | 0.0 [0.0 to 23.2] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 16.8] | 11.1 [1.4 to 34.7]
  Month 30: >=32 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=32 fold rise | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 18.5]
  Month 36: >=4 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=4 fold rise | 0.0 [0.0 to 24.7] | 50.0 [24.7 to 75.3] | 0.0 [0.0 to 16.8] | 50.0 [26.0 to 74.0]
  Month 36: >=8 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=8 fold rise | 0.0 [0.0 to 24.7] | 25.0 [7.3 to 52.4] | 0.0 [0.0 to 16.8] | 38.9 [17.3 to 64.3]
  Month 36: >=16 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=16 fold rise | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 16.8] | 16.7 [3.6 to 41.4]
  Month 36: >=32 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=32 fold rise | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 16.8] | 5.6 [0.1 to 27.3]

58. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Toxin B Specific Antibody Levels at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin B antibodies were measured using neutralization assay.
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 20.6] | 77.8 [52.4 to 93.6] | 0.0 [0.0 to 14.2] | 75.0 [50.9 to 91.3]
  Day 8: >=8 fold rise | 0.0 [0.0 to 20.6] | 55.6 [30.8 to 78.5] | 0.0 [0.0 to 14.2] | 65.0 [40.8 to 84.6]
  Day 8: >=16 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Day 8: >=16 fold rise | 0.0 [0.0 to 20.6] | 33.3 [13.3 to 59.0] | 0.0 [0.0 to 14.2] | 45.0 [23.1 to 68.5]
  Day 8: >=32 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Day 8: >=32 fold rise | 0.0 [0.0 to 20.6] | 33.3 [13.3 to 59.0] | 0.0 [0.0 to 14.2] | 20.0 [5.7 to 43.7]
  Day 30: >=4 fold rise | 0.0 [0.0 to 20.6] | 83.3 [83.3 to 96.4] | 0.0 [0.0 to 14.2] | 90.0 [68.3 to 98.8]
  Day 30: >=8 fold rise | 0.0 [0.0 to 20.6] | 83.3 [58.6 to 96.4] | 0.0 [0.0 to 14.2] | 80.0 [56.3 to 94.3]
  Day 30: >=16 fold rise | 0.0 [0.0 to 20.6] | 55.6 [30.8 to 78.5] | 0.0 [0.0 to 14.2] | 60.0 [36.1 to 80.9]
  Day 30: >=32 fold rise | 0.0 [0.0 to 20.6] | 38.9 [17.3 to 64.3] | 0.0 [0.0 to 14.2] | 45.0 [23.1 to 68.5]
  Month 6: >=4 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=4 fold rise | 6.3 [0.2 to 30.2] | 66.7 [41.0 to 86.7] | 0.0 [0.0 to 14.8] | 70.0 [45.7 to 88.1]
  Month 6: >=8 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=8 fold rise | 0.0 [0.0 to 20.6] | 50.0 [26.0 to 74.0] | 0.0 [0.0 to 14.8] | 55.0 [31.5 to 76.9]
  Month 6: >=16 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=16 fold rise | 0.0 [0.0 to 20.6] | 38.9 [17.3 to 64.3] | 0.0 [0.0 to 14.8] | 35.0 [15.4 to 59.2]
  Month 6: >=32 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=32 fold rise | 0.0 [0.0 to 20.6] | 22.2 [6.4 to 47.6] | 0.0 [0.0 to 14.8] | 25.0 [8.7 to 49.1]
  Month 12: >=4 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=4 fold rise | 12.5 [1.6 to 38.3] | 55.6 [30.8 to 78.5] | 0.0 [0.0 to 16.1] | 50.0 [27.2 to 72.8]
  Month 12: >=8 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=8 fold rise | 0.0 [0.0 to 20.6] | 44.4 [21.5 to 69.2] | 0.0 [0.0 to 16.1] | 50.0 [27.2 to 72.8]
  Month 12: >=16 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=16 fold rise | 0.0 [0.0 to 20.6] | 16.7 [3.6 to 41.4] | 0.0 [0.0 to 16.1] | 20.0 [5.7 to 43.7]
  Month 12: >=32 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=32 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 16.1] | 10.0 [1.2 to 31.7]
  Month 18: >=4 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=4 fold rise | 0.0 [0.0 to 20.6] | 47.1 [23.0 to 72.2] | 5.0 [0.1 to 24.9] | 50.0 [27.2 to 72.8]
  Month 18: >=8 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=8 fold rise | 0.0 [0.0 to 20.6] | 17.6 [3.8 to 43.4] | 0.0 [0.0 to 16.8] | 50.0 [27.2 to 72.8]
  Month 18: >=16 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=16 fold rise | 0.0 [0.0 to 20.6] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 16.8] | 25.0 [8.7 to 49.1]
  Month 18: >=32 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=32 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 15.0 [3.2 to 37.9]
  Month 24: >=4 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=4 fold rise | 6.3 [0.2 to 30.2] | 35.3 [14.2 to 61.7] | 5.0 [0.1 to 24.9] | 47.4 [24.4 to 71.1]
  Month 24: >=8 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=8 fold rise | 6.3 [0.2 to 30.2] | 17.6 [3.8 to 43.4] | 0.0 [0.0 to 16.8] | 26.3 [9.1 to 51.2]
  Month 24: >=16 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=16 fold rise | 0.0 [0.0 to 20.6] | 5.9 [0.1 to 28.7] | 0.0 [0.0 to 16.8] | 15.8 [3.4 to 39.6]
  Month 24: >=32 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=32 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 5.3 [0.1 to 26.0]
  Month 30: >=4 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=4 fold rise | 0.0 [0.0 to 23.2] | 35.3 [14.2 to 61.7] | 0.0 [0.0 to 16.8] | 50.0 [26.0 to 74.0]
  Month 30: >=8 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=8 fold rise | 0.0 [0.0 to 23.2] | 5.9 [0.1 to 28.7] | 0.0 [0.0 to 16.8] | 27.8 [9.7 to 53.5]
  Month 30: >=16 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=16 fold rise | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 5.6 [0.1 to 27.3]
  Month 30: >=32 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=32 fold rise | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 5.6 [0.1 to 27.3]
  Month 36: >=4 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=4 fold rise | 0.0 [0.0 to 24.7] | 31.3 [11.0 to 58.7] | 0.0 [0.0 to 16.8] | 50.0 [26.0 to 74.0]
  Month 36: >=8 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=8 fold rise | 0.0 [0.0 to 24.7] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 16.8] | 38.9 [17.3 to 64.3]
  Month 36: >=16 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=16 fold rise | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 16.8] | 11.1 [1.4 to 34.7]
  Month 36: >=32 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=32 fold rise | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 16.8] | 5.6 [0.1 to 27.3]

59. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Both Toxin A and Toxin B Specific Antibody Levels at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin A and B antibodies were measured using neutralization assay.
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 20
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 20.6] | 72.2 [46.5 to 90.3] | 0.0 [0.0 to 14.2] | 65.0 [40.8 to 84.6]
  Day 8: >=8 fold rise | 0.0 [0.0 to 20.6] | 50.0 [26.0 to 74.0] | 0.0 [0.0 to 14.2] | 50.0 [27.2 to 72.8]
  Day 8: >=16 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Day 8: >=16 fold rise | 0.0 [0.0 to 20.6] | 11.1 [1.4 to 34.7] | 0.0 [0.0 to 14.2] | 35.0 [15.4 to 59.2]
  Day 8: >=32 fold rise | 0.0 [0.0 to 20.6] | 11.1 [1.4 to 34.7] | 0.0 [0.0 to 14.2] | 10.0 [1.2 to 31.7]
  Day 30: >=4 fold rise | 0.0 [0.0 to 20.6] | 83.3 [58.6 to 96.4] | 0.0 [0.0 to 14.2] | 85.0 [62.1 to 96.8]
  Day 30: >=8 fold rise | 0.0 [0.0 to 20.6] | 72.2 [46.5 to 90.3] | 0.0 [0.0 to 14.2] | 70.0 [45.7 to 88.1]
  Day 30: >=16 fold rise | 0.0 [0.0 to 20.6] | 33.3 [13.3 to 59.0] | 0.0 [0.0 to 14.2] | 50.0 [27.2 to 72.8]
  Day 30: >=32 fold rise | 0.0 [0.0 to 20.6] | 16.7 [3.6 to 41.4] | 0.0 [0.0 to 14.2] | 35.0 [15.4 to 59.2]
  Month 6: >=4 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=4 fold rise | 0.0 [0.0 to 20.6] | 55.6 [30.8 to 78.5] | 0.0 [0.0 to 14.8] | 55.0 [31.5 to 76.9]
  Month 6: >=8 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=8 fold rise | 0.0 [0.0 to 20.6] | 38.9 [17.3 to 64.3] | 0.0 [0.0 to 14.8] | 45.0 [23.1 to 68.5]
  Month 6: >=16 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=16 fold rise | 0.0 [0.0 to 20.6] | 16.7 [3.6 to 41.4] | 0.0 [0.0 to 14.8] | 25.0 [8.7 to 49.1]
  Month 6: >=32 fold rise: number analyzed (Participants) | 16 | 18 | 23 | 20
  Month 6: >=32 fold rise | 0.0 [0.0 to 20.6] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 14.8] | 15.0 [3.2 to 37.9]
  Month 12: >=4 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=4 fold rise | 0.0 [0.0 to 20.6] | 44.4 [21.5 to 69.2] | 0.0 [0.0 to 16.1] | 40.0 [19.1 to 63.9]
  Month 12: >=8 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=8 fold rise | 0.0 [0.0 to 20.6] | 27.8 [9.7 to 53.5] | 0.0 [0.0 to 16.1] | 40.0 [19.1 to 63.9]
  Month 12: >=16 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=16 fold rise | 0.0 [0.0 to 20.6] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 16.1] | 10.0 [1.2 to 31.7]
  Month 12: >=32 fold rise: number analyzed (Participants) | 16 | 18 | 21 | 20
  Month 12: >=32 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 16.8]
  Month 18: >=4 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=4 fold rise | 0.0 [0.0 to 20.6] | 47.1 [23.0 to 72.2] | 0.0 [0.0 to 16.8] | 50.0 [27.2 to 72.8]
  Month 18: >=8 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=8 fold rise | 0.0 [0.0 to 20.6] | 29.4 [10.3 to 56.0] | 0.0 [0.0 to 16.8] | 40.0 [19.1 to 63.9]
  Month 18: >=16 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=16 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 10.0 [1.2 to 31.7]
  Month 18: >=32 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 20
  Month 18: >=32 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 16.8]
  Month 24: >=4 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=4 fold rise | 0.0 [0.0 to 20.6] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 16.8] | 36.8 [16.3 to 61.6]
  Month 24: >=8 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=8 fold rise | 0.0 [0.0 to 20.6] | 5.9 [0.1 to 28.7] | 0.0 [0.0 to 16.8] | 15.8 [3.4 to 39.6]
  Month 24: >=16 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=16 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 10.5 [1.3 to 33.1]
  Month 24: >=32 fold rise: number analyzed (Participants) | 16 | 17 | 20 | 19
  Month 24: >=32 fold rise | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 17.6]
  Month 30: >=4 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=4 fold rise | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 33.3 [13.3 to 59.0]
  Month 30: >=8 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=8 fold rise | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 11.1 [1.4 to 34.7]
  Month 30: >=16 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=16 fold rise | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 5.6 [0.1 to 27.3]
  Month 30: >=32 fold rise: number analyzed (Participants) | 14 | 17 | 20 | 18
  Month 30: >=32 fold rise | 0.0 [0.0 to 23.2] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 18.5]
  Month 36: >=4 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=4 fold rise | 0.0 [0.0 to 24.7] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 16.8] | 38.9 [17.3 to 64.3]
  Month 36: >=8 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=8 fold rise | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 16.8] | 27.8 [9.7 to 53.5]
  Month 36: >=16 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=16 fold rise | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 18.5]
  Month 36: >=32 fold rise: number analyzed (Participants) | 13 | 16 | 20 | 18
  Month 36: >=32 fold rise | 0.0 [0.0 to 24.7] | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 18.5]

60. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Toxin A Specific Antibody Levels at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin A antibodies were measured using neutralization assay.
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 7.4] | 75.0 [61.1 to 86.0] | 1.7 [0.0 to 9.2] | 71.2 [57.9 to 82.2]
  Day 8: >=8 fold rise | 0.0 [0.0 to 7.4] | 50.0 [35.8 to 64.2] | 0.0 [0.0 to 6.2] | 55.9 [42.4 to 68.8]
  Day 8: >=16 fold rise | 0.0 [0.0 to 7.4] | 23.1 [12.5 to 36.8] | 0.0 [0.0 to 6.2] | 32.2 [20.6 to 45.6]
  Day 8: >=32 fold rise | 0.0 [0.0 to 7.4] | 13.5 [5.6 to 25.8] | 0.0 [0.0 to 6.2] | 8.5 [2.8 to 18.7]
  Day 30: >=4 fold rise | 0.0 [0.0 to 7.4] | 94.2 [84.1 to 98.8] | 0.0 [0.0 to 6.2] | 84.7 [73.0 to 92.8]
  Day 30: >=8 fold rise | 0.0 [0.0 to 7.4] | 78.8 [65.3 to 88.9] | 0.0 [0.0 to 6.2] | 72.9 [59.7 to 83.6]
  Day 30: >=16 fold rise | 0.0 [0.0 to 7.4] | 67.3 [52.9 to 79.7] | 0.0 [0.0 to 6.2] | 55.9 [42.4 to 68.8]
  Day 30: >=32 fold rise | 0.0 [0.0 to 7.4] | 34.6 [22.0 to 49.1] | 0.0 [0.0 to 6.2] | 32.2 [20.6 to 45.6]
  Month 6: >=4 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=4 fold rise | 0.0 [0.0 to 7.5] | 70.0 [55.4 to 82.1] | 1.8 [0.0 to 9.4] | 61.0 [47.4 to 73.5]
  Month 6: >=8 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=8 fold rise | 0.0 [0.0 to 7.5] | 44.0 [30.0 to 58.7] | 1.8 [0.0 to 9.4] | 39.0 [26.5 to 52.6]
  Month 6: >=16 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=16 fold rise | 0.0 [0.0 to 7.5] | 26.0 [14.6 to 40.3] | 1.8 [0.0 to 9.4] | 18.6 [9.7 to 30.9]
  Month 6: >=32 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=32 fold rise | 0.0 [0.0 to 7.5] | 4.0 [0.5 to 13.7] | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 6.1]
  Month 12: >=4 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=4 fold rise | 0.0 [0.0 to 7.7] | 52.0 [37.4 to 66.3] | 0.0 [0.0 to 6.5] | 36.2 [24.0 to 49.9]
  Month 12: >=8 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=8 fold rise | 0.0 [0.0 to 7.7] | 28.0 [16.2 to 42.5] | 0.0 [0.0 to 6.5] | 24.1 [13.9 to 37.2]
  Month 12: >=16 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=16 fold rise | 0.0 [0.0 to 7.7] | 10.0 [3.3 to 21.8] | 0.0 [0.0 to 6.5] | 5.2 [1.1 to 14.4]
  Month 12: >=32 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=32 fold rise | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 6.2]
  Month 18: >=4 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=4 fold rise | 2.3 [0.1 to 12.0] | 26.5 [14.9 to 41.1] | 0.0 [0.0 to 6.6] | 24.1 [13.9 to 37.2]
  Month 18: >=8 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=8 fold rise | 0.0 [0.0 to 8.0] | 14.3 [5.9 to 27.2] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 6.2]
  Month 18: >=16 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=16 fold rise | 0.0 [0.0 to 8.0] | 2.0 [0.1 to 10.9] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 6.2]
  Month 18: >=32 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=32 fold rise | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 6.2]
  Month 24: >=4 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=4 fold rise | 4.5 [0.6 to 15.5] | 29.2 [17.0 to 44.1] | 9.4 [3.1 to 20.7] | 15.8 [7.5 to 27.9]
  Month 24: >=8 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=8 fold rise | 4.5 [0.6 to 15.5] | 8.3 [2.3 to 20.0] | 5.7 [1.2 to 15.7] | 1.8 [0.0 to 9.4]
  Month 24: >=16 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=16 fold rise | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 6.7] | 1.8 [0.0 to 9.4]
  Month 24: >=32 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=32 fold rise | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 6.3]
  Month 30: >=4 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=4 fold rise | 0.0 [0.0 to 8.6] | 13.3 [5.1 to 26.8] | 0.0 [0.0 to 7.0] | 7.3 [2.0 to 17.6]
  Month 30: >=8 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=8 fold rise | 0.0 [0.0 to 8.6] | 6.7 [1.4 to 18.3] | 0.0 [0.0 to 7.0] | 7.3 [2.0 to 17.6]
  Month 30: >=16 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=16 fold rise | 0.0 [0.0 to 8.6] | 2.2 [0.1 to 11.8] | 0.0 [0.0 to 7.0] | 3.6 [0.4 to 12.5]
  Month 30: >=32 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=32 fold rise | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 6.5]
  Month 36: >=4 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=4 fold rise | 2.4 [0.1 to 12.9] | 18.2 [8.2 to 32.7] | 0.0 [0.0 to 7.1] | 17.0 [8.1 to 29.8]
  Month 36: >=8 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=8 fold rise | 0.0 [0.0 to 8.6] | 2.3 [0.1 to 12.0] | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.1]
  Month 36: >=16 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=16 fold rise | 0.0 [0.0 to 8.6] | 2.3 [0.1 to 12.0] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.7]
  Month 36: >=32 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=32 fold rise | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.7]

61. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Toxin B Specific Antibody Levels at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin B antibodies were measured using neutralization assay.
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 7.4] | 65.4 [50.9 to 78.0] | 0.0 [0.0 to 6.2] | 69.5 [56.1 to 80.8]
  Day 8: >=8 fold rise | 0.0 [0.0 to 7.4] | 48.1 [34.0 to 62.4] | 0.0 [0.0 to 6.2] | 54.2 [40.8 to 67.3]
  Day 8: >=16 fold rise | 0.0 [0.0 to 7.4] | 26.9 [15.6 to 41.0] | 0.0 [0.0 to 6.2] | 37.3 [25.0 to 50.9]
  Day 8: >=32 fold rise | 0.0 [0.0 to 7.4] | 13.5 [5.6 to 25.8] | 0.0 [0.0 to 6.2] | 11.9 [4.9 to 22.9]
  Day 30: >=4 fold rise | 0.0 [0.0 to 7.4] | 80.8 [67.5 to 90.4] | 0.0 [0.0 to 6.2] | 81.4 [69.1 to 90.3]
  Day 30: >=8 fold rise | 0.0 [0.0 to 7.4] | 65.4 [50.9 to 78.0] | 0.0 [0.0 to 6.2] | 64.4 [50.9 to 76.4]
  Day 30: >=16 fold rise | 0.0 [0.0 to 7.4] | 51.9 [37.6 to 66.0] | 0.0 [0.0 to 6.2] | 50.8 [37.5 to 64.1]
  Day 30: >=32 fold rise | 0.0 [0.0 to 7.4] | 34.6 [22.0 to 49.1] | 0.0 [0.0 to 6.2] | 30.5 [19.2 to 43.9]
  Month 6: >=4 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=4 fold rise | 0.0 [0.0 to 7.5] | 64.0 [49.2 to 77.1] | 3.5 [0.4 to 12.1] | 57.6 [44.1 to 70.4]
  Month 6: >=8 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=8 fold rise | 0.0 [0.0 to 7.5] | 38.0 [24.7 to 52.8] | 1.8 [0.0 to 9.4] | 35.6 [23.6 to 49.1]
  Month 6: >=16 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=16 fold rise | 0.0 [0.0 to 7.5] | 22.0 [11.5 to 36.0] | 1.8 [0.0 to 9.4] | 11.9 [4.9 to 22.9]
  Month 6: >=32 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=32 fold rise | 0.0 [0.0 to 7.5] | 12.0 [4.5 to 24.3] | 1.8 [0.0 to 9.7] | 3.4 [0.4 to 11.7]
  Month 12: >=4 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=4 fold rise | 0.0 [0.0 to 7.7] | 46.0 [31.8 to 60.7] | 1.8 [0.0 to 9.7] | 32.8 [21.0 to 46.3]
  Month 12: >=8 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=8 fold rise | 0.0 [0.0 to 7.7] | 30.0 [17.9 to 44.6] | 1.8 [0.0 to 9.7] | 12.1 [5.0 to 23.3]
  Month 12: >=16 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=16 fold rise | 0.0 [0.0 to 7.7] | 14.0 [5.8 to 26.7] | 1.8 [0.0 to 9.7] | 5.2 [1.1 to 14.4]
  Month 12: >=32 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=32 fold rise | 0.0 [0.0 to 7.7] | 4.0 [0.5 to 13.7] | 1.8 [0.0 to 9.7] | 1.7 [0.0 to 9.2]
  Month 18: >=4 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=4 fold rise | 6.8 [1.4 to 18.7] | 32.7 [19.9 to 47.5] | 1.9 [0.0 to 9.9] | 12.1 [5.0 to 23.3]
  Month 18: >=8 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=8 fold rise | 2.3 [0.1 to 12.0] | 20.4 [10.2 to 34.3] | 1.9 [0.0 to 9.9] | 5.2 [1.1 to 14.4]
  Month 18: >=16 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=16 fold rise | 2.3 [0.1 to 12.0] | 4.1 [0.5 to 14.0] | 1.9 [0.0 to 9.9] | 1.7 [0.0 to 9.2]
  Month 18: >=32 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=32 fold rise | 0.0 [0.0 to 8.0] | 2.0 [0.1 to 10.9] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 6.2]
  Month 24: >=4 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=4 fold rise | 20.5 [9.8 to 35.3] | 31.3 [18.7 to 46.3] | 7.5 [2.1 to 18.2] | 12.3 [5.1 to 23.7]
  Month 24: >=8 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=8 fold rise | 13.6 [5.2 to 27.4] | 16.7 [7.5 to 30.2] | 5.7 [1.2 to 15.7] | 5.3 [1.1 to 14.6]
  Month 24: >=16 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=16 fold rise | 9.1 [2.5 to 21.7] | 6.3 [1.3 to 17.2] | 5.7 [1.2 to 15.7] | 1.8 [0.0 to 9.4]
  Month 24: >=32 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=32 fold rise | 6.8 [1.4 to 18.7] | 6.3 [1.3 to 17.2] | 1.9 [0.0 to 10.1] | 0.0 [0.0 to 6.3]
  Month 30: >=4 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=4 fold rise | 7.3 [1.5 to 19.9] | 31.1 [18.2 to 46.6] | 3.9 [0.5 to 13.5] | 18.2 [9.1 to 30.9]
  Month 30: >=8 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=8 fold rise | 4.9 [0.6 to 16.5] | 15.6 [6.5 to 29.5] | 2.0 [0.0 to 10.4] | 7.3 [2.0 to 17.6]
  Month 30: >=16 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=16 fold rise | 2.4 [0.1 to 12.9] | 6.7 [1.4 to 18.3] | 2.0 [0.0 to 10.4] | 3.6 [0.4 to 12.5]
  Month 30: >=32 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=32 fold rise | 2.4 [0.1 to 12.9] | 4.4 [0.5 to 15.1] | 0.0 [0.0 to 7.0] | 1.8 [0.0 to 9.7]
  Month 36: >=4 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=4 fold rise | 9.8 [2.7 to 23.1] | 36.4 [22.4 to 52.2] | 2.0 [0.1 to 10.6] | 13.2 [5.5 to 25.3]
  Month 36: >=8 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=8 fold rise | 4.9 [0.6 to 16.5] | 13.6 [5.2 to 27.4] | 2.0 [0.1 to 10.6] | 1.9 [0.0 to 10.1]
  Month 36: >=16 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=16 fold rise | 4.9 [0.6 to 16.5] | 6.8 [1.4 to 18.7] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.7]
  Month 36: >=32 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=32 fold rise | 2.4 [0.1 to 12.9] | 4.5 [0.6 to 15.5] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.7]

62. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Percentage of Participants Achieving >=4, >=8, >=16 and >=32 Fold Rise From Baseline in Both Toxin A and Toxin B Specific Antibody Levels at Days 8, 30 and Months 6, 12, 18, 24, 30, 36
Description: Toxin A and B antibodies were measured using neutralization assay.
Time Frame: Days 8, 30 and Months 6, 12, 18, 24, 30, 36 after Vaccination 4
Population: as for outcome 43
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 48 | 52 | 58 | 59
percentage of participants
  Day 8: >=4 fold rise | 0.0 [0.0 to 7.4] | 59.6 [45.1 to 73.0] | 0.0 [0.0 to 6.2] | 59.3 [45.7 to 71.9]
  Day 8: >=8 fold rise | 0.0 [0.0 to 7.4] | 34.6 [22.0 to 49.1] | 0.0 [0.0 to 6.2] | 39.0 [26.5 to 52.6]
  Day 8: >=16 fold rise | 0.0 [0.0 to 7.4] | 15.4 [6.9 to 28.1] | 0.0 [0.0 to 6.2] | 18.6 [9.7 to 30.9]
  Day 8: >=32 fold rise | 0.0 [0.0 to 7.4] | 9.6 [3.2 to 21.0] | 0.0 [0.0 to 6.2] | 1.7 [0.0 to 9.1]
  Day 30: >=4 fold rise | 0.0 [0.0 to 7.4] | 78.8 [65.3 to 88.9] | 0.0 [0.0 to 6.2] | 71.2 [57.9 to 82.2]
  Day 30: >=8 fold rise | 0.0 [0.0 to 7.4] | 61.5 [47.0 to 74.7] | 0.0 [0.0 to 6.2] | 55.9 [42.4 to 68.8]
  Day 30: >=16 fold rise | 0.0 [0.0 to 7.4] | 44.2 [30.5 to 58.7] | 0.0 [0.0 to 6.2] | 39.0 [26.5 to 52.6]
  Day 30: >=32 fold rise | 0.0 [0.0 to 7.4] | 19.2 [9.6 to 32.5] | 0.0 [0.0 to 6.2] | 13.6 [6.0 to 25.0]
  Month 6: >=4 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=4 fold rise | 0.0 [0.0 to 7.5] | 54.0 [39.3 to 68.2] | 1.8 [0.0 to 9.4] | 40.7 [28.1 to 54.3]
  Month 6: >=8 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=8 fold rise | 0.0 [0.0 to 7.5] | 26.0 [14.6 to 40.3] | 0.0 [0.0 to 6.3] | 18.6 [9.7 to 30.9]
  Month 6: >=16 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=16 fold rise | 0.0 [0.0 to 7.5] | 14.0 [14.0 to 26.7] | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 6.1]
  Month 6: >=32 fold rise: number analyzed (Participants) | 47 | 50 | 57 | 59
  Month 6: >=32 fold rise | 0.0 [0.0 to 7.5] | 4.0 [0.5 to 13.7] | 0.0 [0.0 to 6.3] | 0.0 [0.0 to 6.1]
  Month 12: >=4 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=4 fold rise | 0.0 [0.0 to 7.7] | 38.0 [24.7 to 52.8] | 0.0 [0.0 to 6.5] | 20.7 [11.2 to 33.4]
  Month 12: >=8 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=8 fold rise | 0.0 [0.0 to 7.7] | 14.0 [5.8 to 26.7] | 0.0 [0.0 to 6.5] | 5.2 [1.1 to 14.4]
  Month 12: >=16 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=16 fold rise | 0.0 [0.0 to 7.7] | 4.0 [0.5 to 13.7] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 6.2]
  Month 12: >=32 fold rise: number analyzed (Participants) | 46 | 50 | 55 | 58
  Month 12: >=32 fold rise | 0.0 [0.0 to 7.7] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.5] | 0.0 [0.0 to 6.2]
  Month 18: >=4 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=4 fold rise | 0.0 [0.0 to 8.0] | 18.4 [8.8 to 32.0] | 0.0 [0.0 to 6.6] | 6.9 [1.9 to 16.7]
  Month 18: >=8 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=8 fold rise | 0.0 [0.0 to 8.0] | 8.2 [2.3 to 19.6] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 6.2]
  Month 18: >=16 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=16 fold rise | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 6.2]
  Month 18: >=32 fold rise: number analyzed (Participants) | 44 | 49 | 54 | 58
  Month 18: >=32 fold rise | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.3] | 0.0 [0.0 to 6.6] | 0.0 [0.0 to 6.2]
  Month 24: >=4 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=4 fold rise | 4.5 [0.6 to 15.5] | 16.7 [7.5 to 30.2] | 3.8 [0.5 to 13.0] | 7.0 [1.9 to 17.0]
  Month 24: >=8 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=8 fold rise | 4.5 [0.6 to 15.5] | 2.1 [0.1 to 11.1] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 6.3]
  Month 24: >=16 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=16 fold rise | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 6.3]
  Month 24: >=32 fold rise: number analyzed (Participants) | 44 | 48 | 53 | 57
  Month 24: >=32 fold rise | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.4] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 6.3]
  Month 30: >=4 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=4 fold rise | 0.0 [0.0 to 8.6] | 4.4 [0.5 to 15.1] | 0.0 [0.0 to 7.0] | 5.5 [1.1 to 15.1]
  Month 30: >=8 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=8 fold rise | 0.0 [0.0 to 8.6] | 2.2 [0.1 to 11.8] | 0.0 [0.0 to 7.0] | 3.6 [0.4 to 12.5]
  Month 30: >=16 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=16 fold rise | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 7.0] | 1.8 [0.0 to 9.7]
  Month 30: >=32 fold rise: number analyzed (Participants) | 41 | 45 | 51 | 55
  Month 30: >=32 fold rise | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 7.9] | 0.0 [0.0 to 7.0] | 0.0 [0.0 to 6.5]
  Month 36: >=4 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=4 fold rise | 2.4 [0.1 to 12.9] | 13.6 [5.2 to 27.4] | 0.0 [0.0 to 7.1] | 3.8 [0.5 to 13.0]
  Month 36: >=8 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=8 fold rise | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.7]
  Month 36: >=16 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=16 fold rise | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.7]
  Month 36: >=32 fold rise: number analyzed (Participants) | 41 | 44 | 50 | 53
  Month 36: >=32 fold rise | 0.0 [0.0 to 8.6] | 0.0 [0.0 to 8.0] | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.7]

63. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Percentage of Participants With Local Reactions by Severity Within 14 Days After Vaccination 4
Description: Local reactions included pain at injection site, swelling and redness collected by using an electronic diary (e-diary). Pain was graded as: mild (grade 1) (did not interfere with activity), moderate (grade 2) (interfered with activity), severe (grade 3) (prevented daily activity) and grade 4 (emergency room visit or hospitalization). Redness and swelling were graded as: mild (2.5-5.0 cm), moderate (>5.0 to 10.0 cm), severe (>10.0 cm) and grade 4 (necrosis). Any local reaction referred to any injection site pain, any swelling, or any redness.
Time Frame: Within 14 days after Vaccination 4
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 22
percentage of participants
  Pain: Any | 6.3 [0.2 to 30.2] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 14.2] | 27.3 [10.7 to 50.2]
  Pain: Mild | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 27.3 [10.7 to 50.2]
  Pain: Moderate | 0.0 [0.0 to 20.6] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Pain: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Pain: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Redness: Any | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 13.6 [2.9 to 34.9]
  Redness: Mild | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 13.6 [2.9 to 34.9]
  Redness: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Redness: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Redness: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Swelling: Any | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 13.6 [2.9 to 34.9]
  Swelling: Mild | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 9.1 [1.1 to 29.2]
  Swelling: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  Swelling: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Swelling: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]

64. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Percentage of Participants With Local Reactions by Severity Within 14 Days After Vaccination 4
Description: as for outcome 63
Time Frame: Within 14 days after Vaccination 4
Population: Safety population: all participants who received at least 1 dose of the investigational product. Here "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 50 | 52 | 58 | 59
percentage of participants
  Pain: Any | 6.0 [1.3 to 16.5] | 23.1 [12.5 to 36.8] | 3.4 [0.4 to 11.9] | 20.3 [11.0 to 32.8]
  Pain: Mild | 6.0 [1.3 to 16.5] | 21.2 [11.1 to 34.7] | 3.4 [0.4 to 11.9] | 16.9 [8.4 to 29.0]
  Pain: Moderate | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 0.0 [0.0 to 6.2] | 3.4 [0.4 to 11.7]
  Pain: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Pain: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Redness: Any | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 0.0 [0.0 to 6.2] | 3.4 [0.4 to 11.7]
  Redness: Mild | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 0.0 [0.0 to 6.2] | 1.7 [0.0 to 9.1]
  Redness: Moderate | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 1.7 [0.0 to 9.1]
  Redness: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Redness: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Swelling: Any | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 0.0 [0.0 to 6.2] | 3.4 [0.4 to 11.7]
  Swelling: Mild | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 0.0 [0.0 to 6.2] | 3.4 [0.4 to 11.7]
  Swelling: Moderate | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Swelling: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Swelling: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]

65. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Percentage of Participants With Systemic Events by Severity Within 14 Days After Vaccination 4
Description: Systemic events included following events: Fever was graded as mild (38.0 to 38.4 degree C), moderate (38.5 to 38.9 degree C), severe (39.0 to 40.0 degree C), grade (G) 4 (>40.0 degree C). Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours), severe (required intravenous hydration)/grade 4 (hospitalization for hypotensive shock). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours), severe (>=6 stools in 24 hours) and G4 (hospitalization). Headache, fatigue, new/worsening muscle pain and new/worsening joint pain was graded as mild (no interference with activity), moderate (some interference with activity), severe (prevents daily activity) and G4 (hospitalization). Any systemic event referred to any fever >= 38.0 degree C, any vomiting, any diarrhea, any headache, any fatigue, any new/worsening muscle pain, or any new or worsening joint pain.
Time Frame: Within 14 days after Vaccination 4
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 22
percentage of participants
  Fever: Any | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 4.2 [0.1 to 21.1] | 0.0 [0.0 to 15.4]
  Fever: Mild | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Fever: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 4.2 [0.1 to 21.1] | 0.0 [0.0 to 15.4]
  Fever: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Fever: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Vomiting: Any | 0.0 [0.0 to 20.6] | 5.6 [0.1 to 27.3] | 4.2 [0.1 to 21.1] | 4.5 [0.1 to 22.8]
  Vomiting: Mild | 0.0 [0.0 to 20.6] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  Vomiting: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 4.2 [0.1 to 21.1] | 0.0 [0.0 to 15.4]
  Vomiting: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Vomiting: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Diarrhea: Any | 12.5 [1.6 to 38.3] | 16.7 [3.6 to 41.4] | 25.0 [9.8 to 46.7] | 13.6 [2.9 to 34.9]
  Diarrhea: Mild | 12.5 [1.6 to 38.3] | 11.1 [1.4 to 34.7] | 12.5 [2.7 to 32.4] | 9.1 [1.1 to 29.2]
  Diarrhea: Moderate | 0.0 [0.0 to 20.6] | 5.6 [0.1 to 27.3] | 4.2 [0.1 to 21.1] | 4.5 [0.1 to 22.8]
  Diarrhea: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 8.3 [1.0 to 27.0] | 0.0 [0.0 to 15.4]
  Diarrhea: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Headache: Any | 6.3 [0.2 to 30.2] | 5.6 [0.1 to 27.3] | 16.7 [4.7 to 37.4] | 9.1 [9.1 to 29.2]
  Headache: Mild | 6.3 [0.2 to 30.2] | 5.6 [0.1 to 27.3] | 8.3 [1.0 to 27.0] | 9.1 [1.1 to 29.2]
  Headache: Moderate | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 8.3 [1.0 to 27.0] | 0.0 [0.0 to 15.4]
  Headache: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Headache: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  Fatigue: Any | 37.5 [15.2 to 64.6] | 27.8 [9.7 to 53.5] | 8.3 [1.0 to 27.0] | 18.2 [5.2 to 40.3]
  Fatigue: Mild | 18.8 [4.0 to 45.6] | 16.7 [3.6 to 41.4] | 4.2 [0.1 to 21.1] | 13.6 [2.9 to 34.9]
  Fatigue: Moderate | 18.8 [4.0 to 45.6] | 11.1 [1.4 to 34.7] | 0.0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  Fatigue: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 4.2 [0.1 to 21.1] | 0.0 [0.0 to 15.4]
  Fatigue: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  New or worsening muscle pain: Any | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 22.7 [7.8 to 45.4]
  New or worsening muscle pain: Mild | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 18.2 [5.2 to 40.3]
  New or worsening muscle pain: Moderate | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  New or worsening muscle pain: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  New or worsening muscle pain: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  New or worsening joint pain: Any | 12.5 [1.6 to 38.3] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  New or worsening joint pain: Mild | 6.3 [0.2 to 30.2] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 14.2] | 4.5 [0.1 to 22.8]
  New or worsening joint pain: Moderate | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  New or worsening joint pain: Severe | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]
  New or worsening joint pain: Grade 4 | 0.0 [0.0 to 20.6] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 14.2] | 0.0 [0.0 to 15.4]

66. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Percentage of Participants With Systemic Events by Severity Within 14 Days After Vaccination 4
Description: as for outcome 65
Time Frame: within 14 days after Vaccination 4
Population: as for outcome 64
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 50 | 52 | 58 | 59
percentage of participants
  Fever: Any | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Fever: Mild | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Fever: Moderate | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Fever: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Fever: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Vomiting: Any | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 3.4 [0.4 to 11.9] | 0.0 [0.0 to 6.1]
  Vomiting: Mild | 0.0 [0.0 to 7.1] | 1.9 [0.0 to 10.3] | 3.4 [0.4 to 11.9] | 0.0 [0.0 to 6.1]
  Vomiting: Moderate | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Vomiting: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Vomiting: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Diarrhea: Any | 16.0 [7.2 to 29.1] | 13.5 [5.6 to 25.8] | 13.8 [6.1 to 25.4] | 11.9 [4.9 to 22.9]
  Diarrhea: Mild | 14.0 [5.8 to 26.7] | 9.6 [3.2 to 21.0] | 8.6 [2.9 to 19.0] | 11.9 [4.9 to 22.9]
  Diarrhea: Moderate | 2.0 [0.1 to 10.6] | 3.8 [0.5 to 13.2] | 5.2 [1.1 to 14.4] | 0.0 [0.0 to 6.1]
  Diarrhea: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Diarrhea: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Headache: Any | 12.0 [4.5 to 24.3] | 9.6 [3.2 to 21.0] | 10.3 [3.9 to 21.2] | 3.4 [0.4 to 11.7]
  Headache: Mild | 8.0 [2.2 to 19.2] | 3.8 [0.5 to 13.2] | 5.2 [1.1 to 14.4] | 1.7 [0.0 to 9.1]
  Headache: Moderate | 4.0 [0.5 to 13.7] | 5.8 [1.2 to 15.9] | 5.2 [1.1 to 14.4] | 1.7 [0.0 to 9.1]
  Headache: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Headache: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  Fatigue: Any | 18.0 [8.6 to 31.4] | 15.4 [6.9 to 28.1] | 24.1 [13.9 to 37.2] | 20.3 [11.0 to 32.8]
  Fatigue: Mild | 12.0 [4.5 to 24.3] | 5.8 [1.2 to 15.9] | 10.3 [3.9 to 21.2] | 11.9 [4.9 to 22.9]
  Fatigue: Moderate | 6.0 [1.3 to 16.5] | 9.6 [3.2 to 21.0] | 10.3 [3.9 to 21.2] | 8.5 [2.8 to 18.7]
  Fatigue: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 3.4 [0.4 to 11.9] | 0.0 [0.0 to 6.1]
  Fatigue: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  New or worsening muscle pain: Any | 6.0 [1.3 to 16.5] | 7.7 [2.1 to 18.5] | 17.2 [8.6 to 29.4] | 6.8 [1.9 to 16.5]
  New or worsening muscle pain: Mild | 4.0 [0.5 to 13.7] | 3.8 [0.5 to 13.2] | 10.3 [3.9 to 21.2] | 1.7 [0.0 to 9.1]
  New or worsening muscle pain: Moderate | 2.0 [0.1 to 10.6] | 3.8 [0.5 to 13.2] | 6.9 [1.9 to 16.7] | 5.1 [1.1 to 14.1]
  New or worsening muscle pain: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  New or worsening muscle pain: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  New or worsening joint pain: Any | 8.0 [2.2 to 19.2] | 3.8 [0.5 to 13.2] | 12.1 [5.0 to 23.3] | 6.8 [1.9 to 16.5]
  New or worsening joint pain: Mild | 4.0 [0.5 to 13.7] | 0.0 [0.0 to 6.8] | 3.4 [0.4 to 11.9] | 1.7 [0.0 to 9.1]
  New or worsening joint pain: Moderate | 4.0 [0.5 to 13.7] | 3.8 [0.5 to 13.2] | 8.6 [2.9 to 19.0] | 5.1 [1.1 to 14.1]
  New or worsening joint pain: Severe | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]
  New or worsening joint pain: Grade 4 | 0.0 [0.0 to 7.1] | 0.0 [0.0 to 6.8] | 0.0 [0.0 to 6.2] | 0.0 [0.0 to 6.1]

67. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Treatment-emergent adverse events are events from dose 4 of study drug to 28 days after dose 4 of study drug that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From Vaccination 4 up to 28 days after Vaccination 4
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 22
Participants | 1 | 0 | 4 | 3

68. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: as for outcome 67
Time Frame: From Vaccination 4 up to 28 days after Vaccination 4
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 51 | 52 | 58 | 59
Participants | 10 | 8 | 17 | 16

69. Secondary Outcome: Extension Stage Day 1, 8 and 30 Regimen: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; lack of efficacy in an approved indication. Treatment-emergent serious adverse events are events from dose 4 of study drug to 6 months after dose 4 of study drug that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From Vaccination 4 up to 6 months after Vaccination 4
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen
Number analyzed (Participants) | 16 | 18 | 24 | 22
Participants | 0 | 0 | 1 | 1

70. Secondary Outcome: Extension Stage Month 0, 1 and 6 Regimen: Number of Participants With Treatment Emergent Serious Adverse Events (SAEs)
Description: as for outcome 69
Time Frame: From Vaccination 4 up to 6 months after Vaccination 4
Population: Safety population: all participants who received at least 1 dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
Number analyzed (Participants) | 51 | 52 | 58 | 59
Participants | 2 | 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: AEs: From Vaccination 1 up to 1 month after Vaccination 3 (up to Month 2 for day regimen and Month 7 for month regimen); from Vaccination 4 up to 36 months (after Vaccination 4) SAEs: From Vaccination 1 through 6 months after Vaccination 3 (Month 7 for day regimen and Month 12 for month regimen); from Vaccination 4 up to 36 months (after Vaccination 4)
Description: SAEs and AEs were grouped by system organ class and preferred term. AEs included AEs collected in the e-diary (local and systemic reactions; systematic assessment) and AEs collected on the case report form at each visit (nonsystematic assessment). Safety population: all participants who received at least 1 dose of the investigational product.
Arm/Group | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen | Placebo: Day 1, 8 and 30 Regimen | Clostridium Difficile Vaccine(100 mcg): Month 0, 1 and 6 Regimen | Clostridium Difficile Vaccine(200 mcg): Month 0, 1 and 6 Regimen | Placebo: Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen
All-Cause Mortality (participants affected / at risk) | 2/182 | 1/184 | 0/61 | 2/183 | 0/183 | 0/61 | 0/16 | 0/18 | 0/24 | 1/22 | 0/51 | 0/52 | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 11/182 | 6/184 | 0/61 | 19/183 | 22/183 | 2/61 | 6/16 | 3/18 | 3/24 | 2/22 | 4/51 | 2/52 | 6/58 | 5/59
Other Adverse Events (participants affected / at risk) | 128/182 | 144/184 | 38/61 | 158/183 | 156/183 | 52/61 | 9/16 | 7/18 | 11/24 | 14/22 | 22/51 | 20/52 | 31/58 | 34/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen (N=182) | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen (N=184) | Placebo: Day 1, 8 and 30 Regimen (N=61) | Clostridium Difficile Vaccine(100 mcg): Month 0, 1 and 6 Regimen (N=183) | Clostridium Difficile Vaccine(200 mcg): Month 0, 1 and 6 Regimen (N=183) | Placebo: Month 0, 1 and 6 Regimen (N=61) | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen (N=16) | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen (N=18) | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen (N=24) | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen (N=22) | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen (N=51) | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen (N=52) | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen (N=58) | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen (N=59)
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Device malfunction (Product Issues) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Meningoencephalitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Chemical burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Carotid artery disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Aortic aneurysm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
B-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clostridium Difficile Vaccine(100 mcg):Day 1, 8 and 30 Regimen (N=182) | Clostridium Difficile Vaccine(200 mcg):Day 1, 8 and 30 Regimen (N=184) | Placebo: Day 1, 8 and 30 Regimen (N=61) | Clostridium Difficile Vaccine(100 mcg): Month 0, 1 and 6 Regimen (N=183) | Clostridium Difficile Vaccine(200 mcg): Month 0, 1 and 6 Regimen (N=183) | Placebo: Month 0, 1 and 6 Regimen (N=61) | 100mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen (N=16) | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen (N=18) | 200mcg Clostridium Difficile Vaccine to Placebo:Day 1, 8 and 30 Regimen (N=24) | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Day 1, 8 and 30 Regimen (N=22) | 100mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen (N=51) | 100mcg Clostridium Difficile Vaccine to 100mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen (N=52) | 200mcg Clostridium Difficile Vaccine to Placebo:Month 0, 1 and 6 Regimen (N=58) | 200mcg Clostridium Difficile Vaccine to 200mcg Clostridium Difficile Vaccine:Month 0,1 and 6 Regimen (N=59)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Retinoschisis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Anorectal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2 | 5 | 4 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Chest pain (General disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Fatigue (General disorders) | 0 | 1 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site bruising (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site erythema (General disorders) | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site haematoma (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site haemorrhage (General disorders) | 9 | 9 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site macule (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site pain (General disorders) | 4 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site pruritus (General disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site swelling (General disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site warmth (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Oedema peripheral (General disorders) | 0 | 2 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pain (General disorders) | 2 | 2 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tenderness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vessel puncture site swelling (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Multiple allergies (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Eye infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Incision site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 6 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Upper respiratory tract infection (Infections and infestations) | 4 | 8 | 2 | 16 | 17 | 5 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Urinary tract infection (Infections and infestations) | 3 | 2 | 0 | 5 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Viral upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 8 | 4 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Root canal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Labyrinthitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Gout (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 6 | 9 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 5 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Headache (Nervous system disorders) | 0 | 2 | 0 | 4 | 6 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Breast calcifications (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Left ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Mitral valve calcification (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Right atrial dilatation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Right ventricular dilatation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Factor V deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypogonadism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Eye disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Glaucoma (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Neovascular age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tooth disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Drug intolerance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site discolouration (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site erosion (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site nodule (General disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Infected bite (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Laryngitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Lenticular injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vitreous injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Blood pressure increased (Investigations) | 0 | 0 | 0 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Fibrin D dimer increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Ophthalmological examination abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Red reflex abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Aortic dilatation (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Breast cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Pyrexia (fever) (General disorders) | 2 | 4 | 0 | 5 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Headache (Nervous system disorders) | 35 | 46 | 16 | 52 | 56 | 23 | 1 | 1 | 4 | 2 | 6 | 5 | 6 | 2 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site erythema (redness) (General disorders) | 10 | 21 | 1 | 11 | 11 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 2 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site pain (pain) (General disorders) | 77 | 92 | 6 | 77 | 83 | 9 | 1 | 1 | 0 | 6 | 3 | 12 | 2 | 12 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Injection site swelling (swelling) (General disorders) | 11 | 19 | 0 | 10 | 16 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 2 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Diarrhoea (diarrhea) (Gastrointestinal disorders) | 26 | 37 | 16 | 65 | 59 | 17 | 2 | 3 | 6 | 3 | 8 | 7 | 8 | 7 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vomiting (Gastrointestinal disorders) | 1 | 5 | 2 | 5 | 4 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Fatigue (General disorders) | 43 | 59 | 20 | 81 | 69 | 24 | 6 | 5 | 2 | 4 | 9 | 8 | 14 | 12 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 15 | 31 | 6 | 35 | 45 | 9 | 2 | 1 | 0 | 1 | 4 | 2 | 7 | 4 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 29 | 41 | 8 | 47 | 42 | 11 | 1 | 0 | 0 | 5 | 3 | 4 | 10 | 4 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Vessel puncture site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Macular cyst (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Allergy to animal (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).
Blood folate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v20.0 was used for coding events till Vaccination 1 to 3 and MedDRA v23.0 was used for coding events Extension Stage (Vaccination 4).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-06-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT02561195/SAP_000.pdf
  • Study Protocol (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT02561195/Prot_001.pdf